IMP : Everolimus

Protocol No.: CRAD001LIC01


Version : 2
Status : Final


# Clinical Development & Medical Affairs

# RAD001, Everolimus

# CRAD001LIC01 / NCT01206764

An Open-Label, Multi-Center Phase 2 Study to Evaluate Everolimus as Monotherapy Treatment for Patients with Metastatic Recurrent and/or Unresectable Renal Cell Carcinoma (EVERMORE)

Trial: Phase II

# RAP Module and appendix deliverables

Author (s)

Document type: RAP

Document status: Final

Release date: 22SEP2017

Number of pages: 101

IMP : Everolimus


Status : Final


# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.



# List of abbreviations used in the text

| ATC | Anatomical Therapeutic Chemical |
|--------|----------------------------------------------|
| AE | Adverse Event |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| BMI | Body Mass Index |
| BUN | Blood Urea Nitrogen |
| CRF | Case Report Form |
| CT | Computerized Tomography |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| ECG | Electrocardiogram |
| GGT | Gamma-Glutamyl-Transferase |
| HDL | High Density Lipoprotein |
| INR | International Normalized Ratio |
| ITT | Intent-to-Treat |
| LDH | Lactate Dehydrogenase |
| LDL | Low Density Lipoprotein |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic Resonance Imaging |
| QC | Quality Control |
| ORR | Objective Response Rate |
| PFS | Progression Free Survival |
| PT | Preferred Term |
| RAP | Reporting Analysis Plan |
| RCC | Renal Cell Carcinoma |
| SAE | Serious Adverse Event |
| SBR | Senior Biostatistical Review |
| SI | Standard International |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| WBC | White Blood Cell |
| WHO | World Health Organization |

IMP : Everolimus

Version : 2 Confidential Protocol No.: CRAD001LIC01 Status : Final 

# **Table of contents**

| 1. | Introduction | ••••• | 6 |
|----|-----------------------------------------------|-------|-----|
| | 1.1 Background and rationale | 6 | |
| | 1.2 Study Description | 6 | |
| 2. | Study Objectives | | 6 |
| | 2.1 Primary | 6 | |
| | 2.2 Secondary | 6 | |
| 3. | Study Design | ••••• | 6 |
| | 3.1 Assessments | 7 | |
| | 3.2 Study Medication | | |
| | 3.3 Treatment Arms | 7 | |
| | 3.4 Randomization and Blinding Procedure | 7 | |
| | 3.5 Sample size calculation | 8 | |
| 4. | Endpoints | | 8 |
| | 4.1 Primary Endpoint | 8 | |
| | 4.1.1 Progression Free Survival Rate | | |
| | 4.2 Secondary Endpoints | 8 | |
| | 4.2.1 Disease Control Rate (SD + PR + CR) | 8 | |
| | 4.2.2 Objective Response Rate and Duration | 8 | |
| | 4.2.3 Overall Survival | 8 | |
| | 4.2.4 Safety Endpoints | 8 | |
| 5. | Analysis Populations | ••••• | 8 |
| 6. | Interim Analysis | | 9 |
| 7. | Statistical Analysis Methods | | 9 |
| | 7.1 General Principles | | |
| | 7.2 Data handling | | |
| | 7.2.1 Calculation of time-to-event | 9 | |
| | 7.2.2 RECIST Criteria | 10 | |
| | 7.2.3 Handling of Missing and Incomplete Data | 10 | |
| | 7.3 Patient Disposition | 13 | |
| | 7.4 Protocol Deviation | 13 | |
| | 7.5 Demographic and Baseline Characteristics | 13 | |
| | 7.6 Time to Event Analysis | 14 | |
| | 7.7 Other Efficacy Analysis | 15 | |
| 8. | Safety Analyses | | .15 |

IMP: Everolimus Version 2 Confidential Protocol No.: CRAD001LIC01 Status Final  8.1 8.2 8.3 8.4 8.5 9. 10. 10.1 10.2 10.3 11.

22SEP2017

Date

**Novartis** 

IMP : Everolimus


Status : Final


#### 1. INTRODUCTION

#### 1.1 Background and rationale

The reporting analysis plan (RAP) is based upon section 10 'Statistical Methods and Data Analysis' of the study protocol. The RAP has been prepared in compliance with ICH E9.

Statistical analyses will be carried out using all available case report form (CRF) data.

#### 1.2 Study Description

This is an open-label, multi-center Phase II study to evaluate RAD001 (everolimus) as monotherapy treatment for patients with metastatic recurrent and/or unresectable renal cell carcinoma (RCC).

The purpose of this study is to demonstrate the safety and efficacy of RAD001, an mTOR inhibitor, as monotherapy in patients with metastatic carcinoma of the kidney who have not received prior systemic treatment, other than cytokine therapy. The proposed dose and schedule (10 mg/day) is based on various Phase 1 and Phase 2 studies (monotherapy and combination therapy) in advanced cancers, including RCC, and a large controlled Phase 3 study (RECORD-1).

Current standard therapies (chemotherapies and cytokine-based therapies) have produced few and short-lived tumor responses, and are associated with severe toxicities. The efficacy of RAD001 as monotherapy in patients who were previously treated with cytokine therapy (Amato et al., 2009), and whose disease had progressed on VEGF-tyrosine kinase inhibitor therapy (Motzer et al., 2008) were recently reported.

# 2. STUDY OBJECTIVES

# 2.1 Primary

The primary objective of the study is to evaluate Progression Free Survival (PFS) rate over time.

# 2.2 Secondary

- 1. To evaluate the disease control rate (stable disease [SD] + partial response [PR] + complete response [CR]) (SD + PR + CR);
- 2. To evaluate the objective response rate (ORR; where ORR = CR + PR);
- 3. To evaluate duration of response;
- 4. To evaluate OS;
- 5. To describe the safety profile of RAD001.

# 3. STUDY DESIGN

This is an open-label, multi-center, single arm Phase II study.

It is anticipated that approximately 142 patients will be enrolled in the study.

The target population is patients with any Memorial Sloan-Kettering Cancer Center prognosis metastatic recurrent and/or unresectable clear cell or non-clear cell carcinoma of the kidney. Patients who have received prior cytokine therapy are permitted to participate in the study.

IMP : Everolimus


Status : Final


#### 3.1 Assessments

Upon provision of written, informed consent patients will be given a unique 9 digit patient number. This will be a combination of their 4 digit center number and 5 digit subject number.

The patient will be assessed for their eligibility to take part in the study (i.e. receive study medication) using the inclusion and exclusion criteria stated in the protocol (Sections 5.1 and 5.2). If the patient fails to start on treatment for any reason, this reason will be entered on the Screening Log. No data for screen failures will be entered into the clinical database.

Patients who are eligible for treatment will be dispensed their study medication on completion of their baseline visit. Patients should present to the clinic on Day 1 and Day 15 of treatment Cycles 1, 2, and 3 and Day 1 of each subsequent treatment cycle to complete the assessments detailed in Table 6 of the protocol, until completion of treatment which will occur when the patient experiences disease progression, unacceptable toxicity, death or discontinues from the study for any other reason. An end of study treatment assessment should then be performed. All patients will have a follow-up visit 28 days after the last dose of the study drug to follow for adverse events (AEs) and serious adverse events (SAEs) that may have occurred after discontinuation from the study.

Tumor response will be assessed at 8 weeks (+/- 1 week), and every 12 weeks (+/- 1 week) thereafter until determination of disease progression and at the end of the study.

Patients who discontinue treatment, or are withdrawn from treatment by the investigator, for any reason, should complete an early discontinuation assessment. All patients who discontinue treatment will continue to have tumor assessments at 12-week intervals until the initiation of new cancer therapy.

The efficacy assessments for this study will be the assessment of tumor response/progression and survival status. Tumor response/progression assessments should be performed by a Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) scan. The same imaging modality used at screening must be used for all subsequent follow-up assessments.

Safety assessments will consist of evaluating AEs and SAEs, laboratory parameters including hematology, chemistry, vital signs and documentation of all concomitant medications and/or therapies. The Karnofsky Performance Status score will also be recorded.

## 3.2 Study Medication

Eligible patients will receive RAD001 (10 mg/day) continuously from Visit 2 (Cycle 1, Day 1) until disease progression, unacceptable toxicity, or death or discontinuation from the study for any other reason. Patients will be instructed to take two 5 mg RAD001 tablets (one tablet after another) orally, with a glass of water at the same time each day, in a fasting state or with a light fat-free meal.

Dose adjustments are permitted in those patients who are unable to tolerate the protocol-specified dosing schedule. Rules for the interruption or modification of dosing are described in Table 2, Table 3 and Table 4 of the protocol.

#### 3.3 Treatment Arms

This is a single arm study with all patients receiving RAD001 (10mg/day). There is no control group for this study.

# 3.4 Randomization and Blinding Procedure

Since this study is an open-label, single arm study no randomization or blinding procedures are required.

IMP : Everolimus


Status : Final


#### 3.5 Sample size calculation

The sample size for this study was determined with reference to estimating a CI for the PFS rate at 10 months, assuming (for simplicity) the use of the normal approximation to the binomial distribution and assuming that a CI for a proportion is based on this normal approximation. To be able to estimate a 95% CI for the PFS rate, centered at 0.50, and having an expected total interval width of approximately 0.27, requires a sample size of 55 patients in each of the 2 cohorts (first- and second-line). With 95% confidence, the expected total interval width is approximately 0.19 for all 110 patients (both cohorts combined).

#### 4. ENDPOINTS

## 4.1 Primary Endpoint

#### 4.1.1 Progression Free Survival Rate

The primary endpoint for this study is progression free survival (PFS). The derivation for this is given in Section 7.2.1.

## 4.2 Secondary Endpoints

# 4.2.1 Disease Control Rate (SD + PR + CR)

Disease control rate is defined in Section 7.2.2.

#### 4.2.2 Objective Response Rate and Duration

Objective response rate and duration are defined in Section 7.2.2.

## 4.2.3 Overall Survival

Overall survival is defined in Section 7.2.1.

#### 4.2.4 Safety Endpoints

The safety endpoints defined for this study are frequency of adverse events and laboratory values.

#### 5. ANALYSIS POPULATIONS

A full description of the patient populations is given below:

Intent-to-treat (ITT) population: Consists of all patients treated with RAD001.

Safety population: Consists of all patients who received at least one dose of the study drug and who have at least one post-baseline safety assessment. Please note that the statement that a patient had no adverse events (on the Adverse Event CRF) constitutes a safety assessment. Patients who have received at least one dose of study drug but who have no post-treatment safety data of any kind would be excluded from the safety population.

The ITT population will be the primary population of interest for the efficacy analyses. The safety population will be used when presenting safety data.

It should also be noted that patients who give informed consent and record any baseline data but are found not to meet the inclusion/exclusion criteria and are not given study medication will be classed as screening failures. No data for these subjects will be recorded in the clinical database. Should a patient receive

IMP : Everolimus


Status : Final


study medication and it is subsequently found that they fail to meet inclusion/exclusion criteria then the patient will be included in the ITT population (and safety if they have at least one post-baseline assessment).

#### 6. INTERIM ANALYSIS

There is no interim analysis planned for this study.

#### 7. STATISTICAL ANALYSIS METHODS

#### 7.1 General Principles

The number of patients in the population of interest will be presented on each table, shown as N=XXX. For data summarized by visit, the N will be the number of patients in the population of interest still present in the study at that visit. See Section 7.3 on Patient Disposition for a full definition.

Data from unscheduled visits will be listed only, except for the End of Treatment row in safety tables if the unscheduled visit is the patient's last on-treatment record.

No visit windowing will be applied for this study. However, it will be checked when summarizing any data that are collected by visit that on-treatment assessments did actually take place prior to the end of treatment date. Should an on-treatment assessment be performed later than the date of last treatment, the data will be listed but will not be included in the summary tables. The timing of off-treatment data will be checked again prior to database lock as data collected within 30 days of end of treatment may be considered valid for use in summary tables in which case this definition will be updated to allow for these cases.

It should be noted this rule does not cover adverse event data which have a separate definition of on-treatment.

## 7.2 Data handling

#### 7.2.1 Calculation of time-to-event

In the following definitions the time of study entry has been defined as date of first dose of study medication (taken from the dosage administration record on the CRF).

The date of last contact (used in the censoring rules below) is collected on the End of Study/Survival Information page of the CRF. However, it should be noted that it is only planned for contact with patients to take place at the clinic visits and so the date of last contact captured on the CRF should always be equal to the date of last visit attended.

#### Progression Free Survival:

PFS is defined as the time from date of first dose of study medication until the date of the first documented disease progression or death due to any cause. Date of progression and date of death will be captured on the CRF.

For the purpose of calculating the PFS Rate if a patient has not progressed or died at the date of analysis cut-off, or when he/she received further anticancer therapy, then their time to progression or death will be censored at the time of last tumor assessment, before the first cut-off date or the anticancer therapy date.

# **Progression Free Survival Rate:**

IMP : Everolimus


Status : Final


The PFS rate is defined as the survival function at the end of the time point based on a Kaplan-Meier analysis of the time to either progression (as per the local radiological review) or death (see next section for handling of censored data).

The time points at which PFS rate will be summarized are: 8 weeks, 20 weeks, 32 weeks, 44 weeks, 56 weeks and every 12 weeks thereafter as appropriate.

#### Overall Survival:

Overall survival is defined as the time fromdate of first dose of study medication until death due to any cause. The date of death will be captured on the CRF.

If a patient is still alive and not lost to follow-up at the end of the study then their time to death will be censored at the date of last contact date, as recorded on the CRF.

If the patient has been lost to follow-up by the end of the study then their time to death will be censored at the date of last contact as recorded on the CRF.

In the event that a date of last contact has not been recorded on the CRF, then the date of the last assessment recorded should be used instead.

## Duration of Response:

The duration of response (CR or PR) is defined as the time from from the first occurrence of PR or CR (as per the local radiological review) until the date of the first documented disease progression or death due to underlying cancer. If a patient has not had an event, duration of response is censored at the date of last adequate tumor assessment prior to starting new anticancer therapy.

# 7.2.2 RECIST Criteria

#### Disease Control Rate:

The disease control rate is based on the data as per local radiological review following the RECIST V1.0 criteria. The disease control rate is defined as the proportion of patients with CR, PR, or SD.

# Objective Response Rate:

The overall tumor response will be based on the data as per local radiological review, following RECIST criteria. The ORR is defined as the proportion of patients with CR or PR.

# 7.2.3 Handling of Missing and Incomplete Data

#### Prior Antineoplastic Therapy:

Missing or partial dates of antineoplastic therapy will be imputed in order to determine the duration of treatment with each therapy. If the end date of antineoplastic therapy is missing or partial the latest possible date will be imputed up until the day prior to start of study medication (since antineoplastic therapy use is pre-study). Partial start dates of antineoplastic therapy will be imputed as the earliest possible date. It should be noted that use of antineoplastic therapy during the study would be considered a protocol deviation. Imputed dates will be for the purpose of calculating duration only and the listing should display only the partial date information recorded on the CRF.

#### Adverse Events (AEs):

In the event of a missing severity for a patient's adverse event, no imputation will be made but this should be raised with Data Management for further discussion since no missing data would be expected for this variable.

IMP : Everolimus


Status : Final


Partial start dates for adverse events will be imputed in order to determine if the event is treatment emergent. The imputation of partial start dates of adverse events will follow the following rules:

| Adverse Event Start Date Imputation | |
|---|---|
| Available Data (YYYY-MM-DD) | Imputation Rule |
| YYYY | If the year part is the same as the year of first dose of study medication, impute with the date of first dose of study medication. |
| | Otherwise, impute with the 1st of January of the known year. |
| YYYY-MM | If the known part is same as the date of first dose of study medication then impute with date of first dose of study medication. |
| | Otherwise, impute with the 1st of the known month. |
| All missing | If the known end date is after date of first dose of study medication then impute with the date of first dose of study medication. |
| | Otherwise, impute with the date of informed consent. |

# Concomitant Medications/Significant Non-Drug Therapies:

Patial start and end dates of medications will be imputed to determine if a medication is concomitant. The imputation of partial start and/or end dates of medications will follow the following rules:


| Medication Start Date | | Medication | n End Date |
|---|---|---|---|
| Available Data | Imputation Rule | Available Data | Imputation Rule |
| (YYYY-MM-DD) | | (YYYY-MM-DD) | |
| YYYY | If the year part is the same as the year of first dose of study medication, impute with the date of first dose of study medication. Otherwise, impute with the 1st of January of the known year. | YYYY | Impute as 31'st December of the known year. |
| YYYY-MM | If the known part is same as the date of first dose of study medication then impute with date of first dose of study medication. | YYYY-MM | Impute as the last day of the known month. |
| | Otherwise, impute with the 1st of the known month. | | |
| All missing | If the known end date is after date of first dose of study medication then impute with the date of first dose of study medication. | All missing | Impute as date of last contact |
| | Otherwise, impute with the date of informed consent. | | |

# **Disease Progression:**

If disease progression or death is documented after one single missing tumor assessment, the actual event date of disease progression/death will be used for the PFS event date. If disease progression is documented after two or more missing tumor assessments, the PFS time of the patient will be censored at the date of the last tumor assessment with overall lesion response of CR, PR or SD.

Additional sensitivity analyses will be performed where:

IMP : Everolimus


Status : Final


1. The actual event date of disease progression/death will be used for the PFS event date, irrespective of whether it is preceded by missing tumor assessments;

2. In case of a documented progression/death after one or more missing tumor assessments, disease progression is considered to have occurred at the next scheduled tumor assessment after the date of the last tumor assessment with overall lesion response of CR, PR, or SD.

# Duration of Response:

The same rules for missing data for calculation of duration of response will be applied as for PFS described above.

### 7.3 Patient Disposition

Patients will be defined as enrolled if they gave written, informed consent to enter the study. Disposition will be assessed at the end of the time of data cut-off for analysis (or at end of treatment if the patient withdraws from the study before then). A patient will be defined as completing treatment if they have not been recorded as discontinuing treatment on the End of Study page of the CRF. If they record any reason for discontinuing treatment on the End of Study page they will be considered as an early withdrawal from treatment. Their primary reason for early discontinuation of treatment will be summarized.

The disposition table will also show the number and percentage of patients in each of the analysis populations and in each stratum (first-line patients and second-line patients). The summaries of safety data that are collected by visit (i.e. laboratory tests and vital signs etc but not adverse events or concomitant medications) will present data relative to the number of patients still present in the study at that visit. A patient will be defined as being still present in the study at Visit X if they have data at Visit X or they have data at a later visit, noting that it cannot be assumed a patient was still in the study at an ontreatment visit if the only later data are from a follow-up visit. A patient with at least one on-treatment visit will be included in the End of Treatment row, even if that one visit is an unscheduled visit.

#### 7.4 Protocol Deviation

Protocol deviations will be identified prior to database lock.

Major protocol deviations will be summarized and tabulated. Other protocol deviations will also be identified, summarized and listed.

#### 7.5 Demographic and Baseline Characteristics

Demographic data including date of birth, sex, race and ethnicity will be collected at Screening Visit 1a. Age will be derived as the age in years at Screening Visit 1a. Age, sex, race, ethnicity, height, weight, BMI and Karnofsky Performance Status will be summarized for the ITT population. In the event of a difference between the safety and ITT populations, this summary of demographic data will be repeated for the safety population.

The date of informed consent, any failed inclusion or exclusion criteria and the source of subject referral will be listed only.

Relevant medical history and current medical conditions are collected at Screening Visit 1a. The number of patients with at least one relevant medical history or current medical condition and at least one active problem will be presented and a summary will also be provided of the medical history by body system and preferred term. These summaries will be performed on the ITT population.

IMP : Everolimus


Status : Final


A pregnancy test is performed at Screening Visit 1a and Baseline Visit 1b and the data collected will be listed only. If any unscheduled pregnancy tests are performed during the treatment or follow-up periods of the study these data will also be listed.

Each patient's prior antineoplastic therapy is recorded at Screening Visit 1a. The number of patients taking each therapy type overall and by setting will be presented along with the total number of separate courses of therapy. Each separate record entered on the CRF will be counted as a separate course of therapy. For each therapy type/setting combination the overall best response per patient will be determined as either Complete Response (best), Partial Response, Stable Disease, Complete Response (unconfirmed), Unknown, Not Applicable or Progressive Disease (worst). The total duration of time per therapy type/setting will be calculated for each patient based on the CRF data. It is expected the duration will be calculated in months and should take into account any overlap in dates recorded on the CRF. See Section 7.2.2 regarding the handling of partial dates. Summaries of prior antineoplastic therapy will be performed on the ITT population, and in the event of a difference between the safety and ITT populations will be repeated for the safety population.

A chest x-ray will be performed at Screening Visit 1a. These data will be summarized presenting the investigator's assessment of abnormality for the safety population.

Data for all chest x-ray assessments throughout the study (including unscheduled) will be listed.

Medications (other than study medication) and significant non-drug therapies used throughout the treatment period are captured on the CRF. These will be coded using the Novartis Drug and Therapy Dictionary (Version Sep 2009). Those that start on or after the first day of dosing with study medication and no later than 30 days after the last dose of study medication, and those that end after the start of study medication (even if started prior to study medication) will be defined as concomitant and will be summarized. Summaries will be presented by Anatomical Therapeutic Classification (ATC) class and preferred term for the safety population. If a patient takes multiple medications/therapies within an ATC class or within an ATC class and preferred term, the patient will be counted once.

#### 7.6 Time to Event Analysis

At each visit where tumor assessment is performed the CRF will capture the RECIST assessment of tumor response according to local radiological review. If disease progression occurs then the End of Treatment pages of the CRF should be completed.

The patient's status at the end of study will be summarized with patients being classed as either alive, dead or lost to follow-up and either having had a relapse/recurrence or not. Further, if the patient has died it will be summarized whether death was due to study indication or not. These summaries will be performed on the ITT population.

The time to event variables are defined in Section 7.2.1.

No statistical test of hypotheses will be performed in this study. PFS rate and 95% confidence intervals will be presented graphically and tabulated, overall and by strata, using the Kaplan-Meier product-limit method. The resulting median PFS will be presented along with 95% CIs. These analyses will be performed on the ITT population.

The analysis of PFS will be repeated for the sensitivity analyses described in Section 7.2.3 and also for Duration of Response.

For Overall Survival the Kaplan-Meier curve will be displayed and the median, 25<sup>th</sup> and 75<sup>th</sup> percentile of the Kaplan-Meier estimate will be reported for the ITT population.

IMP : Everolimus


Status : Final


## 7.7 Other Efficacy Analysis

Disease control rate and ORR (as defined in Section 7.2.2) will be summarized by percentage of subjects along with 95% CIs for the ITT population.

#### 8. SAFETY ANALYSES

All Summaries of safety data will be conducted on the safety population.

#### **8.1 Adverse Events**

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®) Version 12.1 to provide the system organ class (SOC) and preferred term for each AE.

An adverse event will be defined as treatment emergent if it begins on or after the first day of dosing with study medication and no later than 30 days after the last dose of study medication. It is expected that adverse event monitoring will continue for at least 4 weeks after the last dose of study medication but new events occurring after the end of the treatment period will not be recorded on the CRF (unless they are serious or lead to death).

Since adverse events occurring prior to start of study or between signing informed consent and start of study medication should be considered as medical history, it is anticipated that all adverse events will be treatment emergent adverse events. However, in the event of any non-treatment emergent adverse events occurring, these will be indicated on the adverse event listings. Non-treatment emergent adverse events are defined as events that begin prior to the first day of dosing. If these events are Serious Adverse Events (SAEs) then they will also be summarized.

The number of patients experiencing each of the following will be summarized:

- At least one treatment emergent adverse event (TEAE)
- At least one SAE
- At least one SAE with a suspected relationship to study medication
- At least one adverse TEAE event leading to death
- At least one TEAE leading to modification of study medication
- At least one TEAE leading to permanent discontinuation of study medication
- At least one severe TEAE
- At least one TEAE with a suspected relationship to study medication

Serious adverse events will be indicated on the CRF, as will adverse events leading to modification or permanent discontinuation of study medication. The addition of non-drug therapy will not be classed as a modification of study medication.

Adverse events resulting in death are not indicated on the CRF so will be defined as adverse events experienced by a patient who died, with a severity of life-threatening and an end date either missing or equal to the patient's date of death. If a patient has more than one adverse event identified as leading to death then a review by the Novartis medical contact should be performed to determine if each event led to death or whether one supersedes the other (e.g. underlying life threatening condition but patient actually died in an unrelated fatal accident).

All treatment emergent adverse events will be summarized by SOC and preferred term. If a patient experiences multiple events within a SOC the patient will only be counted once within that SOC. If a

IMP : Everolimus


Status : Final


patient experiences multiple preferred terms with in a SOC the patient will be counted for each preferred term but only once for each unique preferred term. Deaths reportable as SAEs and non-fatal SAEs will each be summarized by SOC and preferred term and also listed.

Deaths as reported on the Survival Information and Study Evaluation Completion CRF will be listed.

The handling of missing or partial start and end dates of adverse events, and missing assessments of severity and relationship is covered in Section 7.2.2.

All adverse events captured on the CRF will be listed, regardless of severity, relationship or treatment emergence.

#### 8.2 Cardiac assessments

Standard 12 lead ECG assessments will be performed at the investigator's discretion according to local practice, or if there are signs and symptoms of cardiotoxicity. These data will be listed.

## **8.3 Laboratory Tests**

Each hematology, blood chemistry and serum lipid parameter will be summarized at the Baseline visit (Visit 1a), each cycle, the End of Treatment visit (last assessment up to and including 30 days after last dose date, including unscheduled assessments). The change from baseline will be presented at all post-baseline visits where this can be calculated.

Each coagulation parameter is collected at Screening Visit 1a and Day 1of Cycle 2. These data will be listed.

Each urinalysis parameter will be collected at Screening Visit 1a and subsequently as clinically required. These data will be listed.

The hematology parameters collected are:

White blood cells (WBC), hemoglobin, hematocrit, platelets

**Either:** absolute neutrophils, absolute lymphocytes, absolute eosinophils, absolute basophils and absolute monocytes

**Or:** percentage neutrophils, percentage lymphocytes, percentage eosinophils, percentage basophils and percentage monocytes

The CRF allows for "other" differential counts to be recorded. These results will be listed only.

The blood chemistry parameters collected are:

Urea, blood urea nitrogen, creatinine, lactate dehydrogenase (LDH), total protein, fasting glucose, phosphorus, serum calcium, serum corrected calcium (calculated at baseline only), electrolytes (sodium, magnesium, chloride, and potassium), total bilirubin, gamma-glutamyl-transferase (GGT), albumin, alkaline phosphatase, alanine aminotransferase (ALT) (or SGPT), aspartate aminotransferase (AST) (or SGOT), uric acid

The serum lipid parameters collected are:

Total cholesterol, triglycerides, low-density lipoprotein (LDL), high-density lipoprotein (HDL)

The coagulation parameters collected are:

Prothrombin time (PT), International normalized ratio (INR)

IMP : Everolimus


Status : Final


All laboratory test results will be converted into Standard International (SI) Units by Data Management. Summary tables will present the results in SI Units.

The normal ranges for each parameter will also be included on the database so results can be calculated as being below, within or above the normal range.

Laboratory results will be graded using the Common Toxicity Criteria for Adverse Events (CTCAE) v3.0 document for each parameter where a CTC grade is defined. The parameters with grades defined are:

Hematology: WBC, hemoglobin, platelets and absolute neutrophils

Blood Chemistry: Creatinine, fasting glucose, sodium, magnesium, potassium, albumin, bilirubin, GGT, SGOT (AST), SGPT (ALT) and alkaline phosphatase

Serum Lipid Profile: total cholesterol, triglycerides

A shift table will be presented showing the change from screening to most extreme post-screening value (including the End of Treatment visit and any unscheduled assessments) in CTC grading.

In the event that an unscheduled laboratory test is performed the data from this test will be listed. Unscheduled visit results will only be summarized if the unscheduled visit supersedes the schedules visit's results. I.e. if a scheduled visit is missed, or the laboratory sample is not taken, or there are no results from the laboratory sample, but there is an unscheduled visit occurring prior to the next scheduled visit then the results from the unscheduled visit should be used instead.

# 8.4 Vital Signs

Body temperature, pulse rate, systolic and diastolic blood pressure will be collected at Screening Visit 1a, Baseline Visit 1b, day1 of each cycle and the End of Treatment visit. Height and weight will be collected at Screening Visit 1a only. The vital signs data, including any unscheduled assessments, will be listed.

#### 8.5 Other Safety Assessments

The Karnofsky Performance Status will be assessed at Screening Visit 1a, Baseline Visit 1b, at day 1 of each subsequent cycle and at End of Treatment. The baseline data will be summarized as well as change from baseline for post-baseline visits. All data, including unscheduled assessments, will be listed.

Pulmonary function test (including spirometry, diffusion capacity of carbon monoxide and room air O<sub>2</sub> saturation at rest) will be performed at screening, as medically necessary if there is evidence of non-infectious pneumonitis, and at the end of the study. These data will be listed.

# 8.6 Dosage Administration and Compliance

Study medication, RAD001, is given as a 10mg oral dose to be taken daily until the end of treatment. The dose administered throughout the entire treatment period should be captured on the CRF, including any changes in dosing initiated by the investigator for patients unable to tolerate the planned dosage, and any changes as a result of lack of compliance with the planned dosing regimen by the patient.

The total duration of treatment will be calculated as the number of days from the first to the last dose of study medication inclusive (regardless of any breaks in treatment). The total duration of treatment will also be categorized as up to 4 months, >4 to 8 months, >8 to 12 months, >12 to 16 months, >16 to 20 months, >20 to 24 months and >24 months. This will be calculated by dividing the duration of treatment in days by 365.25/12. The duration in days will be summarized and the number of patients in each 4-month treatment category will also be presented.

All dosage administration data will also be listed.

IMP : Everolimus


Status : Final


# 9. PROGRAMMING/QC PLAN AND SOFTWARE/SYSTEM

All statistical programs will be written in SAS® 9.2 or higher. Programming will be done as per Standard Operating Procedures and Work Instructions. All outputs produced will undergo an independent quality control (QC) and Senior Biostatistical Review (SBR). A QC and SBR Plan will be produced to detail the checks to be performed.

#### 10. TECHNICAL PROGRAMMING SPECIFICATIONS

#### 10.1 General notes

- All data listings should be sorted by country, investigator site, by patient, and by time point within patient, where appropriate.
- Table specific footnotes should be printed below the table, separated from the end of the table by one blank line and left aligned. Avoid numeric references, which can be confused with data; rather use asterisks and other non-numeric symbols to refer to footnotes. Patient-specific footnotes should be avoided.
- For tables that summarize categorical (discrete) data, an Unknown or Missing category should be added to any parameter for which information is not available for any patient. The table should make clear, whether the denominator for percentages includes the Missing category or not.
- Data in columns of a table should be formatted as follows:
- alphanumeric values are left-justified
- whole numbers (e.g., counts) are right-justified
- numbers containing fractional portions are decimal aligned
- All fractional numeric values should be printed with a zero to the left of the decimal point (e.g., 0.12, 0.3). If -0.0 value occurs due to rounding off it should be printed as 0.0.
- Unless otherwise specified, percentage values should be printed with one digit to the right of the decimal point (e.g., 12.8%, 5.4%).
- Less-than-signs "<0.1%" should be printed when values are >0.0 and <0.1%
- If >100% occurs due to rounding off errors then present as 100%
- Missing data should be represented as blank in listings, unless a missing category was explicitly defined.
- Dates should be printed in SAS format DATE9. (e.g. 01Jul1994). Missing portions of dates should be represented on patient listings as dashes (e.g. --Jul1994).

# 10.2 Decimal places

Unless otherwise specified, the estimated mean and median for a set of values should be printed out to one more decimal place than the raw (observed) data and rounded appropriately. Standard errors (or standard deviations) should be printed out to two additional decimal places than the raw (observed) data and rounded appropriately.

IMP : Everolimus


Status : Final


Decimal places for summary tables and listings will be as follows:

- 3 decimal places (p-values; if p-value is less than 0.001, display <0.001).
- data precision + 2 decimal places (standard errors and standard deviations)
- data precision + 1 decimal place (means, medians)
- same as data precision (minimums, maximums)
- 1 decimal place (percentages)
- if percentage =100, no decimal is required.

For example, for age (with raw data in whole years):

| N | XX |
|--------|------|
| Mean | XX.X |
| S.D. | X.XX |
| Min | XX |
| Median | XX.X |
| Max | XX |

#### 10.3 Font size

Font size should be Courier 9 points. Line size is 120 characters. Page size is 30 lines per page.

Column headings should be in initial upper-case characters.

For numeric variables, include "unit" in column heading when appropriate.

#### 11. TABLE AND LISTINGS SHELLS

Each table should be identified by a numeral, and the table designation (e.g., Table 1) should be centered above the title. A decimal system (x.y-c.d) should be used to identify tables and listings with related contents. Tables/listings should be internally paginated in relation to total length (i.e., page number should appear sequentially as page X of N, where N is the total number of pages within a table or listing). The title is in mixed-case characters. The title and table designation are single-spaced, but are separated from the table by at least a double space. The study population or subgroup (e.g., Intent-to-Treat Population) should be identified on the line immediately following the title.

```
Table 14.x-c.d (page n of y)

Title1

Title2

...

TitleN

Population / Subgroup
```

The tables are numbered starting from 14 (as per ICH guidelines), Figures start with 15 and Listings start with 16. Numbering then follows the pattern given below:

```
x takes the values 1 - \text{Baseline (section } 11.1)
```

IMP : Everolimus


Status : Final


2 - Visit (section 11.2)

3 - Lab (section 11.3)

4 – Conmed (section 11.4)

5 - AE/SAE

6 – Time-to-event analysis

c takes the values according to the topics under the respective section x.

d is the unique table number under a topic

# Examples:

The first table under Patient Disposition will be numbered as: Table 14.1-1.1 and Listing 16.1-1.1. Table 14.2-5.3 refers to the third table under Patient Outcome topic in Visit section. See Sections 11.1 to 11.6 for full details of output grouping.

The output should contain information about the program name and the date when output was generated. This information should be given in a footnote (in the bottom row of a page) in the following format:

E:\EMD\EMR62202\abc.sas, (01Jun2003 10:15)

All output should have the four-line header (the 4th line is left blank) indicating the study protocol and the purpose of the analysis at the upper left margin:

**Novartis** 


\_\_\_\_\_\_

# Section 11.1 – Demographic data

This section should include tables and listings for the following data:

- 1. Patient disposition
- 2. Demographic and other baseline characteristics (including medical history)
- 3. Diagnosis and extent of cancer
- 4. Prior antineoplastic therapy
- 5. Chest x-ray

#### Section 11.2 – Visit data

This section should include tables and listings for the following data:

- 1. Vital signs
- 2. Karnofsky Performance status
- 3. Dose administration
- 4. ECG Assessments
- 5. Pulmonary Function Test

## Section 11.3- Lab data

IMP : Everolimus


Status : Final


This section should include tables and listings for the following data:

- 1. Hematology
- 2. Blood Chemistry
- 3. Serum Lipid Parameters
- 4. Coagulation
- 5. Urinalysis

# Section 11.4- Conmed and concomitant diseases data

This section should include tables and listings for the following data:

1. All concomitant medication

# Section 11.5- AE/SAE data

This section should include tables and listings for the following data:

- 1. Summary of all adverse events
- 2. Adverse events by system organ class and preferred term

# Section 11.6- Time-to-event data

This section should include tables and listings for the following data:

- 1. Summary of time to event data
- 2. Survival analysis

IMP : Everolimus


Status : Final


Table of contents for Table, Listing and Figures templates:

Outputs marked with an asterisk will only be produced if the Safety population differs from the ITT population.

| Table Number | Title | Population |
|-----------------|-------------------------------------------|------------|
| Table 14.1-1.1 | Patient Disposition and Analysis | |
| | Populations | |
| Table 14.1-1.2 | Number (%) of Patients with Major | ITT |
| | Protocol Deviations Post Inclusion | |
| Table 14.1-2.1 | Patient Demographic Characteristics | ITT |
| Table 14.1-2.2* | Patient Demographic Characteristics | Safety |
| Table 14.1-2.3 | Diagnosis and Extent of Cancer | ITT |
| Table 14.1-2.4* | Diagnosis and Extent of Cancer | Safety |
| Table 14.1-2.5 | Medical History by System Organ class and | Safety |
| | Preferred Term | |
| Table 14.1-2.6 | Summary Statistics of Change from | Safety |
| | Baseline in Karnofsky Performance Status | |
| Table 14.1-3.1 | Summary of Prior Antineoplastic Therapy | ITT |
| Table 14.1-3.2* | Summary of Prior Antineoplastic Therapy | Safety |
| Table 14.1-3.3 | Duration of Prior Antineoplastic Therapy | ITT |
| | (months) | |
| Table 14.1-3.4* | Duration of Prior Antineoplastic Therapy | Safety |
| | (months) | |
| Table 14.1-5.1 | Summary of Chest X-ray Evaluation at | Safety |
| | Screening | |
| Table 14.2-3.1 | Summary of Duration of Treatment with | Safety |
| | Study Medication | |
| Table 14.3-1.1 | Normal ranges for Hematology and Blood | |
| | Chemistry Parameters | |
| Table 14.3-2.1 | Summary Statistics of Hematology by Visit | Safety |
| Table 14.3-2.2 | Summary Statistics of Change from | Safety |
| | Baseline in Hematology by Visit | |
| Table 14.3-2.3 | Shift Table for CTC Grade for Hematology | Safety |
| | Parameters | |
| Table 14.3-3.1 | Summary Statistics of Blood Chemistry by | Safety |
| | Visit | |
| Table 14.3-3.2 | Summary Statistics of Change from | Safety |
| | Baseline in Blood Chemistry by Visit | |
| Table 14.3-3.3 | Shift Table for CTC Grade for Blood | Safety |
| | Chemistry Parameters | |
| Table 14.3-4.1 | Summary Statistics of Serum Lipid Profile | Safety |
| | by Visit | |
| Table 14.3-4.2 | Summary Statistics of Change from | Safety |

IMP : Everolimus Version: 2 Confidential Protocol No.: CRAD001LIC01 Status : Final

| Page | 23 of 101 |
|------|-----------|
| rage | 25 01 101 |

| | Baseline in Serum Lipid Profile by Visit | |
|---|---|---|
| Table 14.3-4.3 | Shift Table for CTC Grade for Serum Lipid<br>Profile Parameters | Safety |
| Table 14.4-1.1 | Concomitant Medications and Non-Drug Therapies by ATC class and Preferred Term | Safety |
| Table 14.5-1.1 | Summary of Adverse Events | Safety |
| Table 14.5-2.1 | Treatment Emergent Adverse Events by<br>System Organ Class and Preferred Term | Safety |
| Table 14.5-2.2 | Deaths Reportable as Serious Adverse Events by System Organ Class and Preferred Term | Safety |
| Table 14.5-2.3 | Serious Adverse Events by System Organ<br>Class and Preferred Term | Safety |
| Table 14.6-1.1 | Summary of Survival and End of Study<br>Status | ITT |
| Table 14.6-2.1 | Analysis of Progression Free Survival<br>Rate | ITT |
| Table 14.6-2.2 | Analysis of Progression Free Survival<br>Rate – Sensitivity Analysis | ITT |
| Table 14.6-2.3 | Progression Free Survival Descriptive Statistics | ITT |
| Table 14.6-2.4 | Progression Free Survival Descriptive<br>Statistics – Sensitivity Analysis | ITT |
| Table 14.6-2.5 | Duration of Response Descriptive Statistics | ITT |
| Table 14.6-2.6 | Objective Response Rate and Disease Control Rate | ITT |
| Table 14.6-2.7 | Overall Survival Descriptive Statistics | ITT |

IMP : Everolimus


Status : Final


| Figure Number | Title | Population |
|-----------------|----------------------------------------|------------|
| Figure 15.6-2.1 | Kaplan Meier Plot for Progression Free | ITT |
| | Survival | |
| Figure 15.6-2.2 | Kaplan Meier Plot for Progression Free | ITT |
| | Survival – Sensitivity Analysis 1 | |
| Figure 15.6-2.3 | Kaplan Meier Plot for Progression Free | ITT |
| | Survival – Sensitivity Analysis 2 | |
| Figure 15.6-2.4 | Kaplan Meier Plot for Duration of | ITT |
| | Response | |
| Figure 15.6-2.5 | Kaplan Meier Plot for Overall Survival | ITT |


| Listing Number | Title | Population |
|---|---|---|
| Listing 16.1-1.1 | End of Treatment Status | All Treated Patients |
| Listing 16.1-1.2 | Analysis Populations and Strata | All Patients |
| Listing 16.1-1.3 | Failed Inclusion/Exclusion | All Patients |
| | Criteria and Major Protocol | |
| | Deviations | |
| Listing 16.1-1.4 | All Protocol Deviations | All Patients |
| Listing 16.1-2.1 | Patient Demographic | All Patients |
| | Characteristics | |
| Listing 16.1-2.2 | Relevant Medical History/Current | All Patients |
| | Medical Conditions | |
| Listing 16.1-3.1 | Diagnosis and Extent of Cancer | All Patients |
| Listing 16.1-3.2 | Diagnosis and Extent of Cancer – | All Patients |
| | Lesions | |
| Listing 16.1-4.1 | Prior Antineoplastic Therapy – | All Patients |
| | Medication Details | |
| Listing 16.1-4.2 | Prior Antineoplastic Therapy – | All Patients |
| | Response | |
| Listing 16.1-5.1 | Baseline Chest X-Ray Evaluation | All Patients |
| Listing 16.2-1.1 | Vital Signs by Visit | All Treated Patients |
| Listing 16.2-2.1 | Karnofsky Performance Status by | All Treated Patients |
| | Visit | |
| Listing 16.2-3.1 | Study Drug Administration | All Treated Patients |
| Listing 16.2-3.2 | Dosage Administration Details | All Treated Patients |
| Listing 16.2-4.1 | ECG Assessments | All Treated Patients |
| Listing 16.2-5.1 | Pregnancy Test Results | All Patients |
| Listing 16.2-6.1 | Pulmonary Function Test – | All Patients |
| | Spirometry | |
| Listing 16.2-6.2 | Pulmonary Function Test – | All Patients |
| | Diffusion Capacity for Carbon | |
| | Monoxide | |
| Listing 16.2-6.3 | Pulmonary Function Test – Pulse | All Patients |
| | Oximetry | |
| Listing 16.2-7.1 | Post-Baseline Chest X-Ray | All Patients |
| | Evaluation | |
| Listing 16.2-7.2 | Imaging | All Patients |
| Listing 16.3-1.1 | Hematology by Visit | All Treated Patients |
| Listing 16.3-2.1 | Blood Chemistry by Visit | All Treated Patients |
| Listing 16.3-3.1 | Serum Lipid Profile by Visit | All Treated Patients |
| Listing 16.3-4.1 | Coagulation by Visit | All Treated Patients |
| Listing 16.3-5.1 | Urinalysis Dipstick Analysis by<br>Visit | All Treated Patients |
| Listing 16.3-5.2 | Urinalysis Microscopic Analysis<br>by Visit | All Treated Patients |
| Listing 16.4-1.1 | Concomitant Medications and | All Treated Patients |

IMP : Everolimus


Status : Final


| | Non-Drug Therapies | |
|------------------|------------------------------------|----------------------|
| Listing 16.4-2.1 | Antineoplastic Therapy Since | All Treated Patients |
| | Discontinuation of Study Drug | |
| Listing 16.5-1.1 | All Adverse Events | All Treated Patients |
| Listing 16.5-2.1 | Deaths Reportable as SAEs | All Patients |
| Listing 16.5-2.2 | Non-Fatal SAEs | All Patients |
| Listing 16.6-1.1 | <b>RECIST Solid Tumor Response</b> | All Treated Patients |
| | Assessment – Target Lesions | |
| Listing 16.6-1.2 | <b>RECIST Solid Tumor Response</b> | All Treated Patients |
| | Assessment – Non-Target Lesions | |
| Listing 16.6-1.3 | <b>RECIST Solid Tumor Response</b> | All Treated Patients |
| | Assessment – Overall Response | |
| Listing 16.6-1.4 | Survival Status at End of Study | All Treated Patients |
| Listing 16.6-1.5 | Progression and Survival Details | All Treated Patients |
| Listing 16.7-1.1 | Comments Listing | All Patients |

IMP : EverolimusVersion:2Protocol No.: CRAD001LIC01ConfidentialStatus:Final


Table 14.1-1.1 
Patient Disposition and Analysis Populations

| Disposition | Total |
|-----------------------------------------------------|------------|
| Reason | n (%) |
| Enrolled | XX |
| Completed | xx (xx.x%) |
| Withdrawn | xx (xx.x%) |
| Primary reason for early discontinuation of treatme | ent |
| Adverse event(s) | xx (xx.x%) |
| Abnormal laboratory value(s) | xx (xx.x%) |
| Abnormal test procedure result(s) | xx (xx.x%) |
| Patient withdrew consent | xx (xx.x%) |
| Lost to follow-up | xx (xx.x%) |
| Administrative problems | xx (xx.x%) |
| Death | xx (xx.x%) |
| Death due to study indication | xx (xx.x%) |
| Death due to other reason | xx (xx.x%) |
| New cancer therapy | xx (xx.x%) |
| Disease progression | xx (xx.x%) |
| Protocol deviation | xx (xx.x%) |

Percentages are based on the number enrolled in the study. Enrolled is defined as patients who gave informed consent.

Disposition is assessed at the cut off date for analysis therefore completed patients are those remaining on study treatment at this time.

Source: Listings 16.1-1.1 and 16.1-1.2

Programming Note: See Section 7.3 of text for definitions of enrolled, completed and withdrawn.

IMP : Everolimus Version : 2
Protocol No.: CRAD001LIC01 Confidential Status : Final


Table 14.1-1.1 
Patient Disposition and Analysis Populations

| Disposition | Total |
|---------------------------------------------------|------------|
| Reason | n (%) |
| Intent-to-treat population | xx (xx.x%) |
| Safety population | xx (xx.x%) |
| First-line Patients | xx (xx.x%) |
| Second-line Patients | xx (xx.x%) |
| Still present in study at each visit (safety popu | ulation) |
| Baseline Visit | XX |
| Cycle 1 Visit 2 | XX |
| Cycle 1 Visit 3 | XX |
| Cycle 2 Visit 4 | XX |
| Cycle 2 Visit 5 | XX |
| Cycle 3 Visit 6 | XX |
| Cycle 3 Visit 7 | XX |
| Cycle 4 Visit 8 | XX |
| Cycle 5 Visit 9 | XX |
| Cycle 6 Visit 10 | XX |
| Cycle 7 Visit 11 | XX |
| Cycle 8 Visit 12 | XX |
| repeat for all treatment cycles | XX |
| End of Treatment | XX |

Percentages are based on the number enrolled in the study.

A patient is defined as being in the population at a visit if they have data at that visit or a subsequent visit. The population at the End of Treatment visit will be anyone who had data for at least one on-treatment visit.

Source: Listings 16.1-1.1 and 16.1-1.2


| | Total<br>N=xxxx<br>n (%) |
|-----------------------------------------|--------------------------|
| Protocol Deviation Description | |
| Xxxxxxx | xx (xx.x%) |
| Xxxx xxxxx | xx (xx.x%) |
| Xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xx (xx.x%) |
| Etc. | |

Percentages are based on the ITT population. Source: Listing 16.1--1.3


# Table 14.1-2.1  Patient Demographic Characteristics Population ITT

| | Total |
|------------------------------|------------|
| Demographic variable | N=xxxx |
| Age (years) | |
| N N | xx |
| Mean | XX.X |
| SD | xx.xx |
| Min | XX XX |
| Median | XX.X |
| Max | |
| Missing | XX |
| MISSING | XX |
| < 65 years | xx (xx.x%) |
| >= 65 years | xx (xx.x%) |
| , oo yeard | m (m,n) |
| Sex | |
| Male | xx (xx.x%) |
| Female | xx (xx.x%) |
| | , , , , , |
| Race | |
| Caucasian | xx (xx.x%) |
| Black | xx (xx.x%) |
| Oriental | xx (xx.x%) |
| Native American | xx (xx.x%) |
| Pacific Islander | xx (xx.x%) |
| Other | xx (xx.x%) |
| Missing | XX |
| Ethnicity | |
| Hispanic/latino | xx (xx.x%) |
| Chinese | xx (xx.x%) |
| Indian (Indian subcontinent) | xx (xx.x%) |
| Japanese | xx (xx.x%) |
| Mixed ethnicity | xx (xx.x%) |
| Other | xx (xx.x%) |
| Missing | XX |

Demography information is collected at the baseline visit (Visit 1).

Percentages are based on the number of patients in the ITT population with non-missing data for that parameter.

Source: Listing 16.1-2.1, 16.2-1.1 and 16.2-2.1

IMP: Everolimus Version : 2


# Table 14.1-2.1  Patient Demographic Characteristics Population ITT

| | Total |
|----------------------|--------|
| Demographic variable | N=xxxx |
| Height (cm) | |
| N | XX |
| Mean | XX.XX |
| SD | XX.XXX |
| Min | XX.X |
| Median | XX.XX |
| Max | XX.X |
| Missing | xx |
| Weight (kg) | |
| N | XX |
| Mean | XX.XX |
| SD | XX.XXX |
| Min | XX.X |
| Median | XX.XX |
| Max | XX.X |
| Missing | XX |
| BMI (kg/m²) | |
| N | XX |
| Mean | XX.XX |
| SD | XX.XXX |
| Min | XX.X |
| Median | XX.XX |
| Max | XX.X |
| Missing | XX |

Demography information is collected at the screening visit (Visit 1a). Percentages are based on the number of patients in the ITT population with non-missing data for that parameter.

Source: Listing 16.1-2.1, 16.2-1.1 and 16.2-2.1

Programming Note: This table will be repeated for the Safety population if this differs from the ITT population (Table 14.1-2.2).


# Table 14.1-2.1  Patient Demographic Characteristics Population ITT

| | Total |
|------------------------------|------------|
| Demographic variable | N=xxxx |
| Karnofsky Performance Status | |
| 100% | xx (xx.x%) |
| 90% | xx (xx.x%) |
| 80% | xx (xx.x%) |
| 70% | xx (xx.x%) |
| 60% | xx (xx.x%) |
| 50% | xx (xx.x%) |
| 40% | xx (xx.x%) |
| 30% | xx (xx.x%) |
| 20% | xx (xx.x%) |
| 10% | xx (xx.x%) |
| Missing | XX |

Demography information is collected at the screening visit (Visit 1a) for all patients. Percentages are based on the number of patients in the ITT population with non-missing data for that parameter.

Source: Listing 16.1-2.1, 16.2-1.1 and 16.2-2.1

Programming Note: This table will be repeated for the Safety population if this differs from the ITT population (Table 14.1-2.2).


Table 14.1-2.3 
Diagnosis and Extent of Cancer
Population ITT

| | Total |
|-------------------------------------|------------|
| Diagnosis variable | N=xxxx |
| Primary Site of Cancer | |
| Site 1 | xx (xx.x%) |
| Site 2 | xx (xx.x%) |
| Site 3 | xx (xx.x%) |
| | xx (xx.x%) |
| Missing | xx |
| Details of Tumor Histology/Cytology | |
| Histology/Cytology 1 | xx (xx.x%) |
| Histology/Cytology 2 | xx (xx.x%) |
| Histology/Cytology 3 | xx (xx.x%) |
| | xx (xx.x%) |
| Missing | xx |
| Histologic Grade | |
| Well differentiated | xx (xx.x%) |
| Moderately differentiated | xx (xx.x%) |
| Poorly differentiated | xx (xx.x%) |
| Undifferentiated | xx (xx.x%) |
| Unknown | xx (xx.x%) |
| Missing | XX |

Diagnosis and extent of cancer information is collected at the screening visit (Visit 1a). Percentages are based on the number of patients in the ITT population with non-missing data for that parameter.

Source: Listing 16.1-3.1 and 16.1-3.2

Programming Note: This table will be repeated for the Safety population if this differs from the ITT population (Table 14.1-2.4).


# Table 14.1-2.3  Diagnosis and Extent of Cancer Population ITT

| | Total |
|----------------------------------------|--------------------------|
| Diagnosis variable | N=xxxx |
| Stage at Initial Diagnosis | |
| Stage 0 | xx (xx.x%) |
| Stage I | xx (xx.x%) |
| Stage Ia | xx (xx.x%) |
| | xx (xx.x%)<br>xx (xx.x%) |
| Miles Committee | |
| Missing | XX |
| Dosing Phase | |
| Dose escalation phase | xx (xx.x%) |
| Dose expansion phase | xx (xx.x%) |
| Missing | xx |
| Any Target Lesions | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Missing | xx |
| Any Non-Target Lesions | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Missing | XX (XX.XV) |
| 111001119 | AA |
| Any Sites of Metastasis to be Reported | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Missing | XX |

Diagnosis and extent of cancer information is collected at the screening visit (Visit 1a). Percentages are based on the number of patients in the ITT population with non-missing data for that parameter. Source: Listing 16.1-3.1 and 16.1-3.2

Programming Note: This table will be repeated for the Safety population if this differs from the ITT population (Table 14.1-2.4).

IMP : EverolimusVersion:2Protocol No.: CRAD001LIC01ConfidentialStatus:Final


Table 14.1-2.5

Medical History by System Organ Class and Preferred Term
Population Safety

| | Total |
|----------------------------------------------------------|----------------|
| System Organ Class | N = xxxx |
| Preferred Term | n (%) |
| | V - / |
| Any relevant medical history/current medical conditions? | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Any active problems? | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| | (1111 • 11 0 ) |
| System Organ Class 1 | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) |
| Preferred Term 2 | xx (xx.x%) |
| | , , |
| Preferred Term 3 | xx (xx.x%) |
| System Organ Class 2 | xx (xx.x%) |
| Preferred Term 4 | xx (xx.x%) |
| Preferred Term 5 | xx (xx.x%) |

Patients experiencing more than one medical history within a system organ class or within a system organ class and preferred term are only counted once.

Percentages are based on the number of patients in the Safety population.

Source: Listing 16.1-2.2


Table 14.1-2.6 (page 1 of n)
Summary Statistics of Change from Baseline in Karnofsky Performance Status
Population Safety

| | Statistic | | | | | | |
|---|---|---|---|---|---|---|---|
| Visit | n | Missing | Mean | SD | Min | Median | Max |
| Cycle 1 Visit 2 (N=xxxx) | xx | XX | xx.xx | xx.xxx | XX.X | XX.XX | XX.X |
| Cycle 1 Visit 3 (N=xxxx) | xx | xx | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 2 Visit 4 (N=xxxx) | XX | XX | XX.XX | xx.xxx | XX.X | XX.XX | XX.X |
| Cycle 2 Visit 5 (N=xxxx) | XX | XX | XX.XX | xx.xxx | XX.X | XX.XX | XX.X |
| Cycle 3 Visit 6 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 3 Visit 7 (N=xxxx) | XX | XX | XX.XX | xx.xxx | XX.X | XX.XX | XX.X |
| Cycle 4 Visit 8 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 5 Visit 9 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 6 Visit 10 (N=xxxx) | XX | XX | XX.XX | xx.xxx | XX.X | XX.XX | XX.X |
| Cycle 7 Visit 11 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Etc. | | | | | | | |

Programming note: Table continues for remaining Cycles then presents and End of Treatment summary which will be the last on-treatment assessment.


 $\begin{array}{c} \text{Table 14.1-3.1 (page 1 of n)} \\ \text{Summary of Prior Antineoplastic Therapy} \\ \text{Population ITT} \end{array}$ 

| Therapy Type | | Total<br>N=xxxx |
|--------------|---------------------------------|-----------------|
| Setting | Best Response Achieved | n (%) |
| Chemotherapy | | xx (xx.x%) xxx |
| Adjuvant | Overall | xx (xx.x%) |
| | Complete Response | xx (xx.x%) |
| | Partial Response | xx (xx.x%) |
| | Stable Disease | xx (xx.x%) |
| | Complete Response (unconfirmed) | xx (xx.x%) |
| | Unknown | xx (xx.x%) |
| | Not Applicable | xx (xx.x%) |
| | Progressive Disease | xx (xx.x%) |
| Neoadjuvant | Overall | xx (xx.x%) |
| | Complete Response | xx (xx.x%) |
| | Partial Response | xx (xx.x%) |
| | Stable Disease | xx (xx.x%) |
| | Complete Response (unconfirmed) | xx (xx.x%) |
| | Unknown | xx (xx.x%) |
| | Not Applicable | xx (xx.x%) |
| | Progressive Disease | xx (xx.x%) |

Percentages of patients on each therapy type/setting combination are based on the ITT population. Patients are counted once under the best response level achieved within that therapy type/setting combination and percentages are based on the number of patients receiving that therapy type/setting combination.

Source: Listing 16.1-4.1

Programming Note: Table continues for the Chemotherapy/Therapeutic, Chemotherapy/Prevention and then for the therapy types Hormonal Therapy, Immunotherapy, Targeted Therapy and Other Therapy.

This table will be repeated for the Safety population if this differs from the ITT population (Table 14.1-3.2).


### Table 14.1-3.3 (page 1 of n) Duration of Prior Antineoplastic Therapy (months) Population ITT

| N=xxxx<br>n (%) |
|-----------------|
| n (%) |
| xx (xx.x%) |
| xx (xx.x%) |
| XX |
| XX.X |
| XX.XX |
| XX.X |
| xx |
| xx (xx.x%) |
| XX |
| XX.X |
| XX.XX |
| XX.X |
| XX |

Percentages of patients on each therapy type/setting combination are based on the ITT population. Source: Listing 16.1-4.1

Programming Note: Table continues for the Chemotherapy/Therapeutic, Chemotherapy/Prevention and then for the therapy types Hormonal Therapy, Immunotherapy, Targeted Therapy and Other Therapy. This table will be repeated for the Safety population if this differs from the ITT population (Table 14.1-3.4).


Table 14.1-5.1
Summary of Chest X-ray Evaluation at Screening
Population Safety

| Description | Total<br>N = xxxx<br>n (%) |
|--------------------------------------|----------------------------|
| X-ray interpretation | |
| Number with assessment | XX |
| Normal | xx (xx.x%) |
| Clinically insignificant abnormality | xx (xx.x%) |
| Clinically significant abnormality | xx (xx.x%) |
| Missing | XX |

Percentages are based on the number of patients in the Safety population who had the relevant assessment performed.

Source: Listings 16.1-5.1


Table 14.2-3.1 
Summary of Duration of Treatment with Study Medication
Population Safety

| | Total |
|------------------|------------|
| | N = xxxx |
| Overall (days) | |
| N | XX |
| Min | XX |
| Median | XX.X |
| Max | XX |
| Missing | XX |
| >0 to 4 months | xx (xx.x%) |
| >4 to 8 months | xx (xx.x%) |
| >8 to 12 months | xx (xx.x%) |
| >12 to 16 months | xx (xx.x%) |
| >16 to 20 months | xx (xx.x%) |
| >20 to 24 months | xx (xx.x%) |
| >24 months | xx (xx.x%) |

Percentages are based on the number of patients in the Safety Population. Source: Listing 16.2-3.1


| Parameter | Unit | Lab Number | Gender | Age Range | Lower Limit | Upper Limit |
|---|---|---|---|---|---|---|
| xxxxxxxxxxx | xx | xxxxx | Male | xx-xx | xx | xx |
| | | | | xx-xx | XX | XX |
| | | | Female | xx-xx | XX | XX |
| | | | | xx-xx | XX | XX |
| | | xxxxx | Male | | XX | XX |
| | | | Female | | XX | XX |
| xxxxxxxxxx | xx | xxxxx | Male | | xx | xx |
| | | | Female | | XX | XX |

. . .

Programming Note: Will need to confirm once ranges are available - if ranges are in SI units and hence do not vary across lab then the "lab number" column can be dropped.


### Table 14.3-2.1 (page 1 of n) Summary Statistics of Hematology by Visit Population Safety

| - | | | | Statistic | | | |
|---|---|---|---|---|---|---|---|
| Visit | n | Missing | Mean | SD | Min | Median | Max |
| Parameter: WBC (units) | | | | | | | |
| Baseline (N=xxxx) | XX | XX | XX.XX | XX.XXX | xx.x | XX.XX | XX.X |
| Cycle 1 Visit 2 (N=xxxx) | XX | XX | XX.XX | XX.XXX | xx.x | XX.XX | XX.X |
| Cycle 1 Visit 3 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 2 Visit 4 (N=xxxx) | XX | xx | XX.XX | XX.XXX | XX.X | XX.XX | xx.x |
| Cycle 2 Visit 5 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 3 Visit 6 (N=xxxx) | XX | xx | XX.XX | XX.XXX | XX.X | XX.XX | xx.x |
| Cycle 3 Visit 7 (N=xxxx) | xx | xx | XX.XX | XX.XXX | XX.X | XX.XX | xx.x |
| Cycle 4 Visit 8 (N=xxxx) | xx | xx | XX.XX | XX.XXX | XX.X | XX.XX | xx.x |
| Cycle 5 Visit 9 (N=xxxx) | xx | XX | XX.XX | XX.XXX | XX.X | xx.xx | xx.x |
| Etc. | | | | | | | |
| End of Treatment (N=xxxx) | XX | xx | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |

Source: Listing 16.3-1.1

Programming note: Table continues for all Cycles. Repeat for each hematology parameter in turn noting that absolute and percentage differentials need to be summarized separately. Results should be shown in SI units.


| | | | | Statistic | | | |
|---|---|---|---|---|---|---|---|
| Visit | n | Missing | Mean | SD | Min | Median | Max |
| Parameter: WBC (units) | | | | | | | |
| Cycle 1 Visit 2 (N=xxxx) | xx | XX | xx.xx | xx.xx | xx.x | XX.XX | XX.X |
| Cycle 1 Visit 3 (N=xxxx) | XX | XX | XX.XX | xx.xxx | xx.x | XX.XX | XX.X |
| Cycle 2 Visit 4 (N=xxxx) | XX | XX | xx.xx | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 2 Visit 5 (N=xxxx) | XX | XX | xx.xx | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 3 Visit 6 (N=xxxx) | XX | XX | xx.xx | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 3 Visit 7 (N=xxxx) | xx | XX | xx.xx | XX.XXX | XX.X | XX.XX | xx.x |
| Cycle 4 Visit 8 (N=xxxx) | xx | xx | xx.xx | XX.XXX | xx.x | XX.XX | xx.x |
| Cycle 5 Visit 9 (N=xxxx) | xx | xx | xx.xx | XX.XXX | xx.x | XX.XX | xx.x |
| Cycle 6 Visit 10 (N=xxxx) | xx | XX | xx.xx | xx.xxx | XX.X | xx.xx | xx.x |
| Cycle 7 Visit 11 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | XX.XX | XX.X |
| Etc. | | | | | | | |

Source: Listing 16.3-1.1

Programming note: Table continues for all Cycles, then presents an End of Treatment summary which will be the last ontreatment assessment. Repeat for each hematology parameter in turn noting that absolute and percentage differentials need to be summarized separately. Results should be shown in SI units.


Table 14.3-2.3 (page 1 of n)
Shift Table for CTC Grade for Hematology Parameters
Population Safety

| | | Screening Visit la (N=xxxx) | | | | | |
|---|---|---|---|---|---|---|---|
| | | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Total | Missing |
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n |
| Parameter: WBC (units) | | | | | | | |
| Most Extreme Post-<br>Screening Visit 1a Value<br>(N=xxxx) | Grade 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Grade 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (100%) | Xx |
| | Missing | Xx | Xx | Xx | Xx | XX | Xx |
| Parameter: Hemoglobin (units) | | | | | | | |
| Most Extreme Post-<br>Screening Visit 1a Value<br>(N=xxxx) | Grade 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Grade 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | Xx |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (100%) | Xx |
| | Missing | XX | XX | XX | XX | XX | XX |
| Etc. | | | | | | | |

CTC grades are calculated from V3.0 of the CTCAE manual.

Percentages are based on the number of patients in the Safety Population with data at Screening and the visit of interest.

Source: Listing 16.3-1.1

Programming Note: Repeat for each hematology parameter for those parameters that have a CTC grade defined (see SAP text).


### Table 14.3-3.1 (page 1 of n) Summary Statistics of Blood Chemistry by Visit Population Safety

| | | | | Statistic | | | |
|---|---|---|---|---|---|---|---|
| Visit | n | Missing | Mean | SD | Min | Median | Max |
| Parameter: Urea (units) | | | | | | | |
| Baseline (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 1 Visit 2 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 1 Visit 3 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 2 Visit 4 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 2 Visit 5 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 3 Visit 6 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 3 Visit 7 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 4 Visit 8 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 5 Visit 9 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 6 Visit 10 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 7 Visit 11 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Etc. | | | | | | | |

Source: Listing 16.3-2.1

Programming note: Table continues for remaining Cycles then presents and End of Treatment summary which will be the last on-treatment assessment. Repeat for each blood chemistry parameter in turn. Results should be shown in SI units.


| | Statistic | | | | | | |
|---|---|---|---|---|---|---|---|
| Visit | n | Missing | Mean | SD | Min | Median | Max |
| Parameter: Urea (units) | | | | | | | |
| Cycle 1 Visit 2 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 1 Visit 3 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 2 Visit 4 (N=xxxx) | xx | XX | XX.XX | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 2 Visit 5 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 3 Visit 6 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 3 Visit 7 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 4 Visit 8 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 5 Visit 9 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 6 Visit 10 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 7 Visit 11 (N=xxxx) | xx | XX | xx.xx | xx.xxx | XX.X | xx.xx | xx.x |
| Etc. | | | | | | | |

Source: Listing 16.3-2.1

Programming note: Table continues for remaining Cycles then presents and End of Treatment summary which will be the last on-treatment assessment. Repeat for each blood chemistry parameter in turn. Results should be shown in SI units.


# $\begin{array}{c} \text{Table 14.3-3.3 (page 1 of n)} \\ \text{Shift Table for CTC Grade for Blood Chemistry Parameters} \\ \text{Population Safety} \end{array}$

| | | | Screen | ning Visit 1a | (N=xxxx) | | |
|---|---|---|---|---|---|---|---|
| | | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Total | Missing |
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n |
| Parameter: Creatinine (un. | its) | | | | | | |
| Most Extreme Post-<br>Screening Visit 1a Value<br>(N=xxxx) | Grade 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (100%) | XX |
| | Missing | XX | Xx | Xx | Xx | XX | XX |
| Parameter: Fasting Glucose | e (units) | | | | | | |
| Most Extreme Post-<br>Screening Visit 1a Value<br>(N=xxxx) | Grade 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx |
| | Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (100%) | XX |
| | Missing | XX | Xx | Xx | Xx | XX | XX |
| Etc. | | | | | | | |

CTC grades are calculated from V3.0 of the CTCAE manual.

Percentages are based on the number of patients in the Safety Population with data at Screening and the visit of interest.

Source: Listing 16.3-2.1

Programming Note: Repeat for each blood chemistry parameter that has a CTC grade defined (see SAP text).


## Table 14.3-4.1 (page 1 of n) Summary Statistics of Serum Lipid Profile by Visit Population Safety

| - | | | | Statistic | | | |
|---|---|---|---|---|---|---|---|
| Visit | n | Missing | Mean | SD | Min | Median | Max |
| Parameter: Total Cholesterol | (units) | | | | | | |
| Baseline (N=xxxx) | XX | XX | xx.xx | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 1 Visit 2 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 1 Visit 3 (N=xxxx) | xx | XX | xx.xx | XX.XXX | XX.X | XX.XX | xx.x |
| Cycle 2 Visit 4 (N=xxxx) | xx | XX | xx.xx | XX.XXX | XX.X | XX.XX | xx.x |
| Cycle 2 Visit 5 (N=xxxx) | xx | XX | xx.xx | XX.XXX | XX.X | XX.XX | xx.x |
| Cycle 3 Visit 6 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 3 Visit 7 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 4 Visit 8 (N=xxxx) | XX | XX | xx.xx | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 5 Visit 9 (N=xxxx) | XX | XX | XX.XX | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 6 Visit 10 (N=xxxx) | XX | XX | xx.xx | XX.XXX | XX.X | XX.XX | XX.X |
| Cycle 7 Visit 11 (N=xxxx) | XX | XX | xx.xx | XX.XXX | XX.X | XX.XX | XX.X |
| Etc. | | | | | | | |

Source: Listing 16.3-3.1

Programming note: Table continues for remaining Cycles then presents and End of Treatment summary which will be the last on-treatment assessment. Repeat for each blood chemistry parameter in turn. Results should be shown in SI units.


| | | | | Statistic | | | |
|---|---|---|---|---|---|---|---|
| Visit | n | Missing | Mean | SD | Min | Median | Max |
| Parameter: Total Cholesterol ( | units) | | | | | | |
| Cycle 1 Visit 2 (N=xxxx) | XX | XX | XX.XX | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 1 Visit 3 (N=xxxx) | xx | XX | XX.XX | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 2 Visit 4 (N=xxxx) | XX | XX | XX.XX | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 2 Visit 5 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 3 Visit 6 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 3 Visit 7 (N=xxxx) | xx | XX | XX.XX | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 4 Visit 8 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 5 Visit 9 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 6 Visit 10 (N=xxxx) | xx | XX | xx.xx | xx.xxx | xx.x | xx.xx | xx.x |
| Cycle 7 Visit 11 (N=xxxx) | xx | XX | xx.xx | XX.XXX | XX.X | XX.XX | xx.x |
| Etc. | | | | | | | |

Source: Listing 16.3-3.1

Programming note: Table continues for remaining Cycles then presents and End of Treatment summary which will be the last on-treatment assessment. Repeat for each serum lipid profile parameter in turn. Results should be shown in SI units.


 $\begin{array}{c} \text{Table 14.3-4.3 } \\ \text{Shift Table for CTC Grade for Serum Lipid Profile Parameters} \\ \text{Population Safety} \end{array}$ 

| | | Screening Visit 1a (N=xxxx) | | | | | |
|---|---|---|---|---|---|---|---|
| | | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Total | Missing |
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n |
| Parameter: Total Choleste | rol (units) | | | | | | |
| Most Extreme Post-<br>Screening Visit 1a Value<br>(N=xxxx) | Grade 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx |
| | Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (100%) | XX |
| | Missing | xx | xx | xx | xx | XX | XX |
| Parameter: Triglycerides | (units) | | | | | | |
| Most Extreme Post-<br>Screening Visit 1a Value<br>(N=xxxx) | Grade 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx |
| | Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Grade 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX |
| | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (100%) | XX |
| | Missing | XX | XX | XX | XX | XX | XX |

CTC grades are calculated from V3.0 of the CTCAE manual.

Percentages are based on the number of patients in the Safety Population with data at Screening and the visit of interest.

Source: Listing 16.3-3.1

Novartis 22SEP2017 Date


Protocol No.: CRAD001LIC01 Confidential : Final Status

> 

Table 14.4-1.1 (page 1 of n) Concomitant Medications and Non-Drug Therapies by ATC class and Preferred Term Population Safety

| ATC Class | Total<br>N = xxxx |
|------------------|-------------------|
| Preferred Term | n (%) |
| ATC Class 1 | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) |
| Preferred Term 2 | xx (xx.x%) |
| Preferred Term 3 | xx (xx.x%) |
| ATC Class 2 | xx (xx.x%) |
| Preferred Term 4 | xx (xx.x%) |
| Preferred Term 5 | xx (xx.x%) |

Patients receiving more than one medication/therapy within an ATC Class or within an ATC Class and preferred term are only counted once.

Percentages are based on the number of patients in the Safety population.

Source: Listing 16.4-1.1


Table 14.5-1.1 
Summary of Adverse Events
Population Safety

| Events | Total<br>N = xxxx<br>n (%) |
|---|---|
| At least one treatment emergent adverse event | xx (xx.x%) |
| At least one serious adverse event<br>At least one adverse event leading to death | xx (xx.x%)<br>xx (xx.x%) |
| At least one adverse event leading to discontinuation of study medication At least one adverse event leading to modification of study medication | xx (xx.x%)<br>xx (xx.x%) |
| At least one severe adverse event<br>At least one adverse event with suspected relationship to study medication | xx (xx.x%)<br>xx (xx.x%) |

Percentages are based on the number of patients in safety population. Source: Listings 16.5-1.1


| | Total |
|---------------------------------------|------------|
| System Organ Class | N = xxxx |
| Preferred Term | n (%) |
| All treatment emergent adverse events | xx (xx.x%) |
| SOC 1 | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) |
| Preferred Term 2 | xx (xx.x%) |
| Preferred Term 3 | xx (xx.x%) |
| SOC 2 | xx (xx.x%) |
| Preferred Term 4 | xx (xx.x%) |
| Preferred Term 5 | xx (xx.x%) |
| Eta | |
| Etc. | |

Patients are counted once within each System Organ Class and Preferred Term or once within each System Organ Class for the summary row.

Percentages are based on the number of patients in safety population.

The table is sorted by system organ class then preferred term within system organ class alphabetically. Source: Listing 16.5-1.1

Programming Note: Use same template for the following tables (but with different source listings).

- Table 14.5-2.2 Deaths Reportable as Serious Adverse Events by System Organ Class and Preferred Term
- Table 14.5-2.3 Serious Adverse Events by System Organ Class and Preferred Term


#### 

| | | Total<br>N = xxxx<br>n (%) |
|---|---|---|
| Alive at end of study | Overall<br>With recurrence | xx (xx.x%)<br>xx (xx.x%) |
| Died | Without recurrence Overall | xx (xx.x%)<br>xx (xx.x%) |
| Died due be shudu indicabies | Due to study indication Due to other reason | xx (xx.xx)<br>xx (xx.xx) |
| Died due to study indication Died due to other reason | Already experienced recurrence No recurrence Already experienced recurrence | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Lost to follow-up | No recurrence Overall | xx (xx.x%)<br>xx (xx.x%) |
| 1000 00 10110 up | Already experienced recurrence<br>No recurrence | xx (xx.x%)<br>xx (xx.x%) |

Percentages are based on the number of patients in ITT population. With recurrence refers to subjects that had disease progression prior to death. Source: Listings 16.6-1.2 and 16.6-1.4


### Table 14.6-2.1  Analysis of Progression Free Survival Rate Population ITT

| | First-line Patients | Second-line Patients | Total |
|---|---|---|---|
| | N = xxxx | N = xxxx | N = xxxx |
| PFS Events | xxx | xxx | xxx |
| PFS Rate | xx.xx | xx.xx | xx.xx |
| 95% CI for PFS Rate | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |

Number of patients achieving PFS = number of subject that experienced progression or died prior to the time of data analysis cut-off.

PFS Rate = survival function at the time of data analysis cut-off based on a Kaplan-Meier analysis of time to either progression or death.

The 95% CI also comes from the Kaplan-Meier analysis.

Source: Listings 16.6-1.5


#### 

| | First-line Patients $N = xxxx$ | Second-line Patients $N = xxxx$ | $\begin{array}{ccc} \text{Total} \\ \text{N} = \text{xxxx} \end{array}$ |
|---|---|---|---|
| Sensitivity Analysis 1: | | | |
| PFS Events | xxx | xxx | xxx |
| PFS Rate | XX.XX | XX.XX | XX.XX |
| 95% CI for PFS Rate | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |
| Sensitivity Analysis 2: | | | |
| PFS Events | xxx | xxx | xxx |
| PFS Rate | XX.XX | XX.XX | XX.XX |
| 95% CI for PFS Rate | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |

Number of patients achieving PFS = number of subject that experienced progression or died prior to the time of data analysis cut-off.

PFS Rate = survival function at the time of data analysis cut-off based on a Kaplan-Meier analysis of time to either progression or death.

The 95% CI also comes from the Kaplan-Meier analysis.

Sensitivity Analysis 1 = Actual event date of disease progression/death used for the PFS event date, regardless of whether is it proceeded by missing tumor assessments.

Sensitivity Analysis 2 = In case of a documented progression/death after one of more missing tumor assessments, disease progression is considered to have occurred at the next scheduled tumor assessment after the date of last tumor assessment with overall lesion response of CR, PR, or SD.

Source: Listings 16.6-1.5


### Table 14.6-2.3  Progression Free Survival Descriptive Statistics Population ITT

| | | | Product Limit Estimates | | | |
|---|---|---|---|---|---|---|
| | | | Survival | 95% CI of | Failure | Survival |
| Time to Event | Censored * | Event # | Rate | Survival Rate | Rate | Standard Error |
| <= Week 8 | XX | xx | x.xxxx | (x.xxxx-x.xxxx) | x.xxxx | x.xxxx |
| <=Week 20 | XX | XX | X.XXXX | (x.xxxx-x.xxxx) | X.XXXX | X.XXXX |
| <=Week 32 | XX | XX | X.XXXX | (x.xxxx-x.xxxx) | X.XXXX | X.XXXX |
| <=Week 44 | XX | XX | X.XXXX | (x.xxxx-x.xxxx) | x.xxxx | x.xxxx |
| <=Week 56 | XX | XX | x.xxxx | (x.xxxx-x.xxxx) | x.xxxx | X.XXXX |
| Etc. | | | | | | |

Source: Listings 16.6-1.5

Programming Note: Table continues for every 12 week assessment as appropriate until analysis data cut-off.

 $<sup>\</sup>star$  Censored is defined as the number of patients who have discontinued from the study for any reason other than progression/death within the time period.

<sup>#</sup> Event is progression/death within the time period.


Protocol No.: CRAD001LIC01 Confidential : Final Status

> 

#### Table 14.6-2.3  Progression Free Survival Descriptive Statistics Population ITT

| | Total |
|-------------------|----------------|
| | N = xxxx |
| Median (95% CI) | xx.xx (xx.xxx) |
| Number Assessed | XX |
| Number Censored | XX |
| Number Uncensored | XX |

Source: Listings 16.6-1.5

Programming Note: Use previous template for the following tables. - Table 14.6-2.5 Duration of Response Descriptive Statistics - Population ITT


Table 14.6-2.4 (page 1 of 4)
Progression Free Survival Descriptive Statistics - Sensitivity Analysis
Population ITT

| | | | Product Limit Estimates | | | |
|---|---|---|---|---|---|---|
| | | | Survival | 95% CI of | Failure | Survival |
| Time to Event | Censored * | Event # | Rate | Survival Rate | Rate | Standard Error |
| Sensitivity Analysis 1: | | | | | | |
| <= Week 8 | XX | XX | X.XXXX | (x.xxxx-x.xxxx) | X.XXXX | x.xxxx |
| <=Week 20 | XX | XX | X.XXXX | (x.xxxx-x.xxxx) | X.XXXX | X.XXXX |
| <=Week 32 | XX | XX | X.XXXX | (x.xxxx-x.xxxx) | X.XXXX | X.XXXX |
| <=Week 44 | XX | XX | X.XXXX | (x.xxxx-x.xxxx) | X.XXXX | x.xxxx |
| <=Week 56 | XX | XX | X.XXXX | (x.xxxx-x.xxxx) | X.XXXX | X.XXXX |
| Etc. | | | | | | |

Sensitivity Analysis 1 = Actual event date of disease progression/death used for the PFS event date, regardless of whether is it proceeded by missing tumor assessments.

Sensitivity Analysis 2 = In case of a documented progression/death after one of more missing tumor assessments, disease progression is considered to have occurred at the next scheduled tumor assessment after the date of last tumor assessment with overall lesion response of CR, PR, or SD.

Source: Listings 16.6-1.5

Programming Note: Table continues for every 12 week assessment as appropriate until analysis data cut-off.

 $<sup>\</sup>star$  Censored is defined as the number of patients who have discontinued from the study for any reason other than progression/death within the time period.

<sup>#</sup> Event is progression/death within the time period.


### Table 14.6-2.4 (page 2 of 4) Progression Free Survival Descriptive Statistics - Sensitivity Analysis Population ITT

| | Total |
|-------------------|----------------|
| | N = xxxx |
| Sensitivity 1: | |
| Median (95% CI) | xx.xx (xx.xxx) |
| Number Assessed | XX |
| Number Censored | XX |
| Number Uncensored | XX |

Sensitivity Analysis 1 = Actual event date of disease progression/death used for the PFS event date, regardless of whether is it proceeded by missing tumor assessments.

Sensitivity Analysis 2 = In case of a documented progression/death after one of more missing tumor assessments, disease progression is considered to have occurred at the next scheduled tumor assessment after the date of last tumor assessment with overall lesion response of CR, PR, or SD.

Source: Listings 16.6-1.5

Programming Note: Repeat for Sensitivity Analysis 2


Table 14.6-2.6 
Objective Response Rate and Disease Control Rate
Population ITT

| | Total |
|------------------------------------|-------------|
| | N = xxxx |
| Objective Response | |
| Patients with CR, n (%) | xx (xx.x%) |
| Patients with PR, n (%) | xx (xx.x%) |
| Objective Response Rate, n (%) | xx (xx.x%) |
| 95% CI for Objective Response Rate | xx.x - xx.x |
| Disease Control | |
| Patients with CR, n (%) | xx (xx.x%) |
| Patients with PR, n (%) | xx (xx.x%) |
| Patients with SD, n (%) | xx (xx.x%) |
| Disease Control Rate, n (%) | xx (xx.x%) |
| 95% CI for Disease Control Rate | xx.x - xx.x |

Source: Listings 16.6-1.5


# Table 14.6-2.7  Overall Survival Descriptive Statistics Population ITT

| | Total<br>N = xxxx |
|--------------------------|------------------------|
| 25th Percentile (95% CI) | xx.xx (xx.xxx, xx.xxx) |
| Median (95% CI) | xx.xx (xx.xxx, xx.xxx) |
| 75th Percentile (95% CI) | xx.xx (xx.xxx, xx.xxx) |
| Number Assessed | xx |
| Number Censored | XX |
| Number Uncensored | XX |

Source: Listings 16.6-1.5


Figure 15.6-2.1 
Kaplan Meier Plot for Progression Free Survival
Population ITT




Programming Note: Use same template for the following figures.

- Figure 15.6-2.2 Kaplan Meier Plot for Progression Free Survival Sensitivity Analysis 1, Population ITT
- Figure 15.6-2.3 Kaplan Meier Plot for Progression Free Survival Sensitivity Analysis 2, Population ITT
- Figure 15.6-2.4 Kaplan Meier Plot for Duration of Response, Population ITT
- Figure 15.6-2.5 Kaplan Meier Plot for Overall Survival, Population ITT


Listing 16.1-1.1 (page 1 of n)
End of Treatment Status
All Treated Patients

| Country/<br>Centre/<br>Patient | Date/Day of<br>Last Dose | Status at<br>Time of<br>Analysis | Reason for Not Completing Treatment<br>Period | Follow-Up for<br>Post-<br>Treatment<br>Evaluations? | Follow-Up<br>for<br>Survival? |
|---|---|---|---|---|---|
| Xxxxxxxxxx/ | ddmmmyyyy/ | Completed | | Yes | No |
| Xxxx-xxxxx<br>Xxxxxxxxxx/ | Xx<br>ddmmmyyyy/ | Discontinued | New cancer therapy | Yes | Yes |
| Xxxx-xxxxx<br>Xxxxxxxxxx/ | Xx<br>ddmmmyyyy/ | Discontinued | Protocol deviation - | Yes | Yes |
| Xxxx-xxxxx | xx | | xxxxxxxxxxxxxxxx | | |

Day is calculated relative to the day of first dose of study medication. These data are collected at the end of the treatment period.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier.


Listing 16.1-1.2 (page 1 of n)
Analysis Populations and Strata
All Patients

| Country/<br>Centre/<br>Patient | Date of<br>Informed<br>Consent | <pre>Intent-to-Treat Population?</pre> | Safety Population? | Strata |
|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | ddmmmyyyy | Yes/No | Yes/No | First-line |
| XXXXXXXXXX<br>XXXXXXXXXXX/<br>XXXX-XXXXX | ddmmmyyyy | Yes/No | Yes/No | Second-line |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | ddmmmyyyy | Yes/No | Yes/No | First-line |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier.


Listing 16.1-1.3 (page 1 of n)
Failed Inclusion/Exclusion Criteria and Major Protocol Deviations
All Patients

| Country/<br>Centre/<br>Patient | Inclusion/Exclusion Criteria Not Met | Major Protocol Deviations Post-Inclusion |
|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx<br>Xxxxxxxxxx/<br>Xxxx-xxxxx<br>Xxxxxxxxxx/ | Xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | *************************************** |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Only list patients who have either failed an inclusion/exclusion criteria and/or had a major protocol deviation post-inclusion.


Listing 16.1-1.4 (page 1 of n)
All Protocol Deviations
All Patients

| Country/<br>Centre/<br>Patient | Deviation Code | Date of Deviation<br>(Day) | Deviation Description | Comment |
|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx<br>Xxxxxxxxx/<br>Xxxx-xxxxx<br>Xxxxxxxxxx/<br>Xxxx-xxxxx | XXX | ddmmmyyyy (xx)/ | Xxxxxxxxxxxx | xxxxxxxxxxxxx |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier.


Listing 16.1-2.1 (page 1 of n)
Patient Demographic Characteristics
All Patients

| Country/<br>Centre/<br>Patient | Date of<br>Birth /<br>Age (years) | Sex | Race | Ethnicity | Child Bearing Potential? | Source of Referral |
|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | ddmmmyyyy / | Male | Caucasian | | | ER or hospital |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | ddmmmyyyy / | Female | Black | | Able to bear children | Radio advertisement |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | ddmmmyyyy /<br>xx | Female | Oriental | Japanese | Post-menopausal | Friend/family member |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier.


### Listing 16.1-2.2 (page 1 of n) Relevant Medical History/Current Medical Conditions All Patients

| Country/<br>Centre/<br>Patient | System Organ Class/<br>Preferred Term/<br>History/Condition | Date of Diagnosis/<br>Surgery | Active Problem? |
|---|---|---|---|
| Xxxxxxxxxx/ | Xxxxxxxxxxxxxx/ | ddmmmyyyy | Yes/No |
| Xxxx-xxxx | Xxxxxxxxxxxxxxxx/ | | |
| | Xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | |
| Xxxxxxxxxx/ | Xxxxxxxxxxxxxxxxx/ | ddmmmyyyy | Yes/No |
| Xxxx-xxxx | Xxxxxxxxxxxxxxx/ | | |
| | Xxxxxxxxxxxxxxxxxxxxxxx | | |
| Xxxxxxxxxx/ | Xxxxxxxxxxxxxxxxxxxx/ | ddmmmyyyy | Yes/No |
| Xxxx-xxxx | Xxxxxxxxxxxxxxxxxxxx/ | | |
| | xxxxxxxxxxx | | |
| | xxxxxxxxxxxx | | |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Conditions should be ordered by date of diagnosis/surgery with oldest condition shown first.


Listing 16.1-3.1 (page 1 of n)
Diagnosis and Extent of Cancer
All Patients

| Country/<br>Centre/<br>Patient | Primary Site<br>of Cancer | Tumor<br>Histology/<br>Cytology | Histologic<br>Grade | Date of<br>Initial<br>Diagnosis | Stage at<br>Initial<br>Diagnosis | Date of<br>First<br>Recurrence/<br>Relapse | Date of<br>Most Recent<br>Recurrence/<br>Relapse | Dosing<br>Phase |
|---|---|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Xxxxxxxxxxx | Xxxxxxxxxx | Xxxxxxxxxx | ddmmmyyyy | Xxxxx | ddmmmyyyy | ddmmmyyyy | Xxxxxx |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Xxxxxxxxxx | Xxxxxxxxx | Xxxxxxxxxx | ddmmmyyyy | Xxxxxx | ddmmmyyyy | ddmmmyyyy | Xxxxxxxx |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Xxxxxxxxxx | Xxxxxxxx | Xxxxxxxxxx | ddmmmyyyy | Xxxxxx | ddmmmyyyy | ddmmmyyyy | xxxxxxx |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier.


Listing 16.1-3.2 (page 1 of n)
Diagnosis and Extent of Cancer - Lesions
All Patients

| Country/<br>Centre/<br>Patient | Any Target<br>Lesions? | Any Non-<br>Target<br>Lesions? | Any Sites of Metastasis? | Metastatic<br>Site(s) |
|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Yes | Yes | Yes | Xxxxxxxxx |
| | | | | Xxxxxxxxxx<br>Xxxxxxxxxx |
| | | | | Xxxxxxxxxx |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Yes | Yes | No | |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | No | Yes | No | |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Metastatic sites should be ordered by the order they appear in the CRF.


## Listing 16.1-4.1 (page 1 of n) Prior Antineoplastic Therapy - Medication Details All Patients

| Country/<br>Centre/<br>Patient | Regimen<br>Number | Therapy Type<br>(Number of<br>Cycles) | Medicatio<br>n | First Dose<br>Date (Day)<br>/Last Dose<br>Date (Day) | Duration<br>of<br>Therapy<br>(months) | Cumulative<br>Dose (Unit) | Planned<br>Dose<br>(Unit) | Route | Setting |
|---|---|---|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Chemotherapy (xx) | xxxxxxxxx | ddmmmyyyy (xx)/ ddmmmyyyy (xx) | xxx | xx (Unit) | xx<br>(Unit) | xx | Therapeutic |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Immunotherapy<br>(xx) | xxxxxxxxx | ddmmmyyyy (xx)/ ddmmmyyyy (xx) | xxx | xx (Unit) | xx<br>(Unit) | xx | Adjuvant |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Other:<br>xxxxxxxx (xx) | xxxxxxxx | ddmmmyyyy (xx)/ ddmmmyyyy (xx) | xxx | xx (Unit) | xx<br>(Unit) | xx | Prevention |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Therapy should be ordered by Regimen Number.


Listing 16.1-4.2 (page 1 of n)
Prior Antineoplastic Therapy - Response
All Patients

| Country/<br>Centre/ Patient | Regimen<br>Number | Therapy Type | Medication | Best<br>Response | Date of<br>Best<br>Response | Duration<br>of<br>Response<br>(Months) | Reason for<br>Discontinuation<br>of Therapy | Date of<br>Progression |
|---|---|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Chemotherapy | xxxxxxxxx | Complete<br>Response | ddmmmyyyy | xx | Adverse event(s) | |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Immunotherapy | xxxxxxxxx | Partial<br>Response | ddmmmyyyy | XX | Disease<br>Progression | ddmmmyyyy |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Other:<br>xxxxxxxx | xxxxxxxx | Unknown | ddmmmyyyy | xx | Other: xxxxxxxx | |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Therapy should be ordered by Regimen Number. If necessary the Best Response column should use abbreviations as follows: CR=complete response, PR=partial response, SD=stable disease, PD=progressive disease, CRU=complete response, unconfirmed, UNK=unknown, NA=not applicable and these abbreviations should be footnoted.


Listing 16.1-5.1 (page 1 of n)
Baseline Chest X-Ray Evaluation
All Patients

| Country/<br>Centre/<br>Patient | Chest X-Ray<br>Performed? | Chest X-Ray<br>Date/<br>Day | Interpretation | Clinically Significant<br>Abnormalities |
|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Yes/No | ddmmmyyyy/<br>xx | Normal | |
| <pre></pre> | Yes/No | ddmmmyyyy/<br>xx | Clinically insignificant abnormality | |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Yes/No | ddmmmyyyy/<br>xx | Clinically significant abnormality | Xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Multiple clinically significant abnormality details should be listed in the order they appear on the CRF.


Listing 16.2-1.1 (page 1 of n)
Vital Signs by Visit
All Treated Patients

| Country/<br>Centre/ | | Assessment | Height | BMI | Weight | Body<br>Temperature | Sitting<br>Pulse | Sitting Blood<br>Pressure (bpm) | |
|---|---|---|---|---|---|---|---|---|---|
| Patient Visit | Date/Day | (cm) | $(kg/m^2)$ | (kg) | (°C) | (bpm) | Systolic | Diastolic | |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening<br>Visit la | ddmmmyyyy/<br>xx | xxx | xxx | xxx | xx.x | xxx | xxx | xxx |
| AAAA AAAAA | Baseline<br>Visit 1b | ddmmmyyyy/<br>xx | | | | XX.X | XXX | xxx | xxx |
| | Cycle 1<br>Visit 2 | ddmmmyyyy/<br>xx | | | | XX.X | xxx | XXX | xxx |
| | Cycle 2<br>Visit 4 | ddmmmyyyy/<br>xx | | | | XX.X | XXX | xxx | Xxx |
| | Cycle 3<br>Visit 6 | ddmmmyyyy/<br>xx | | | | XX.X | XXX | XXX | XXX |

Day is calculated relative to the day of first dose of study medication.

IMP: Everolimus Version : 2


Listing 16.2-2.1 (page 1 of n)
Karnofsky Performance Status by Visit
All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Assessment<br>Date/Day | Performance Status |
|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit 1a | ddmmmyyyy/<br>xx | 100%: Normal, no complaints |
| | Baseline Visit 1b | ddmmmyyyy/<br>xx | 90%: Able to carry on normal activity, minor signs or symptoms of disease |
| | Cycle 1 Visit 2 | ddmmmyyyy/<br>xx | 90%: Able to carry on normal activity, minor signs or symptoms of disease |
| | Cycle 2 Visit 4 | ddmmmyyyy/<br>xx | 80%: Normal activity with effort; some signs or symptoms of disease |
| | Cycle 3 Visit 6 | ddmmmyyyy/<br>xx | 90%: Able to carry on normal activity, minor signs or symptoms of disease |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then by visit date. There is no date of assessment on the CRF page where unscheduled assessments are captured so these assessments cannot be slotted into the correct date order. Therefore unscheduled assessments for a patient will appear at the end of the listing and a footnote will be added regarding this.


Listing 16.2-3.1 (page 1 of n) Study Drug Administration All Treated Patients

| Country/ | | | |
|-------------|---------------|--------------|------------------|
| Centre/ | Start Date of | | Total Daily Dose |
| Patient | Study Drug | Planned Dose | Administered |
| Xxxxxxxxxx/ | ddmmmyyyy | xxxx | XXXX |
| Xxxx-xxxxx | | | |


Listing 16.2-3.2 (page 1 of n)
Dosage Administration Details
All Treated Patients

| Country/<br>Centre/<br>Patient | Regimen<br>Number | Planned<br>Dose (mg) | Actual<br>Dose (mg) | Regimen | Dose<br>Change? | Reason for<br>Change | Start<br>Date/Day | End<br>Date/Day |
|---|---|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 01 | 10 | 10 | o.d/q.d. | No | Lab Test<br>Abnormality | ddmmmyyyy/ | ddmmmyyyy/ |
| AAAA AAAAA | 02 | 10 | 5 | o.d/q.d. | Yes | nonormaticy | ddmmmyyyy/<br>xx | ddmmmyyyy/<br>xx |
| | 03 | 10 | 10 | o.d/q.d. | No | | ddmmmyyyy/<br>xx | ddmmmyyyy/<br>xx |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then by visit date. It may be necessary to present Reason For Change using the following abbreviations: AE=adverse event, DOS=dosing error, LAB=lab test abnormality, SCH=scheduling conflict, DIS=dispensing error. If so, these abbreviations will be footnoted.


Listing 16.2-4.1 (page 1 of n) ECG Assessments All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Assessment<br>Date/Day | Result |
|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit la | ddmmmyyyy/<br>xx | Normal |
| | Baseline Visit 1b | ddmmmyyyy/<br>xx | Clinically Significant Abnormality: xxxxxxxxxxx |
| | Cycle 1 Visit 2 | ddmmmyyyy/<br>xx | Normal |
| | Cycle 2 Visit 4 | ddmmmyyyy/<br>xx | Normal |
| | Cycle 3 Visit 6 | ddmmmyyyy/<br>xx | Clinically Insignificant Abnormality |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Any unscheduled assessments should be included and labeled "Unscheduled Visit". ECG assessments are only performed at the investigator's discretion, only records where the ECG was performed will be presented.


Listing 16.2-5.1 (page 1 of n)
Pregnancy Test Results
All Patients

| Country/<br>Centre/ | 771 - 1 h | Carrala Data (Dan | Paralle |
|---|---|---|---|
| Patient | Visit | Sample Date/Day | Result |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Baseline Visit 1b | ddmmmyyyy/ xx | Negative/Positive |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Baseline Visit 1b | ddmmmyyyy/ xx | Negative/Positive |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Baseline Visit 1b | ddmmmyyyy/ xx | Negative/Positive |
| | Unscheduled Visit | ddmmmyyyy/ xx | Negative/Positive |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Only female patients need to be included on the listing.


Listing 16.2-6.1 (page 1 of n)
Pulmonary Function Test - Spirometry
All Patients

| Country/<br>Centre/<br>Patient | Visit | Test<br>Date/Day | Total Lung<br>Capacity (L) | Forced Vital<br>Capacity (L) | Forced Expiratory Volume in One Second (L) | Functional<br>Residual<br>Capacity (L) | Residual<br>Capacity (L) |
|---|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening<br>Visit la<br>End of<br>Treatment | ddmmmyyyy/<br>xx<br>ddmmmyyyy/<br>xx | x.x<br>x.x | x.x<br>x.x | x.x<br>x.x | x.x<br>x.x | x.x<br>x.x |

Day is calculated relative to the day of first dose of study medication.


Listing 16.2-6.2 (page 1 of n) Pulmonary Function Test  $\,$  - Diffusion Capacity for Carbon Monoxide All Patients

| Country/<br>Centre/<br>Patient | Visit | Was DLCO<br>Done? | Test<br>Date/Day | Diffusion<br>Capacity for CO | Unit |
|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening<br>Visit la | Yes | ddmmmyyyy/<br>xx | xx.xx | xxxxxxxxx |
| | End of<br>Treatment | No | | | |

Day is calculated relative to the day of first dose of study medication.


Listing 16.2-6.3 (page 1 of n)
Pulmonary Function Test - Pulse Oximetry
All Patients

| Country/<br>Centre/<br>Patient | Visit | Was Pulse<br>Oximetry<br>Done? | Test<br>Date/Day | Functional<br>Residual<br>Capacity (%) |
|---|---|---|---|---|
| Xxxxxxxxx/<br>Xxxx-xxxxx | Screening<br>Visit la<br>End of<br>Treatment | Yes<br>No | ddmmmyyyy/<br>xx | xxx |

Day is calculated relative to the day of first dose of study medication.


Listing 16.2-7.1 (page 1 of n)
Post-Baseline Chest X-Ray Evaluation
All Patients

| Country/<br>Centre/<br>Patient | Visit | Chest X-Ray<br>Performed? | Chest X-<br>Ray Date/<br>Day | Interpretation | Clinically<br>Significant<br>Abnormalities | Abnormality<br>Compared to<br>Baseline |
|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Cycle 4<br>Visit 8 | Yes/No | ddmmmyyyy/<br>xx | Normal | | |
| | | Yes/No | ddmmmyyyy/<br>xx | Clinically insignificant abnormality | | |
| | | Yes/No | ddmmmyyyy/<br>xx | Clinically significant abnormality | Xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | New or worsened |
| | | | | | xxxxxxxxxxxxxxxx | Not compared<br>Unchanged |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier and visit date. Multiple clinically significant abnormality details should be listed in the order they appear on the CRF.


Listing 16.2-7.2 (page 1 of n)

Imaging

All Patients

| Country/<br>Centre/<br>Patient | Visit | Date of<br>Scan/Day | Scan Category | Location/ Site | Scan Type | Findings |
|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening<br>Visit la | ddmmmyyyy/<br>xx | Chest, Abdomen and Pelvis | Other: xxxxxxx | CT scan (with contrasts) | xxxxxx |
| | | ddmmmyyyy/<br>xx | Brain | Other: xxxxxxxx | CT scan (with contrasts) | xxxxxx |
| | | ddmmmyyyy/<br>xx | Bone | Bone | | xxxxxxx |
| | ••• | | | | | |

Day is calculated relative to the day of first dose of study medication.


Listing 16.3-1.1 (page 1 of n)
Hematology by Visit
All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Sample<br>Date/ Day | Laboratory<br>Number / Name | Parameter | Result<br>(units) | CTC Grade |
|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit | ddmmmyyyy/<br>xx | Xxxxxxxxxxx/<br>xxxxxxx | WBC | xx (unit) | Xx |
| | | | | Hemoglobin | xx (unit) | Xx |
| | | | | Platelets | xx (unit) | Xx |
| | | | | Hematocrit | xx (unit) | |
| | | | | Neutrophils | xx (unit) | Xx |
| | | | | Lymphocytes | xx (unit) L | |
| | | | | Eosinophils | xx (unit) | |
| | | | | Basophils | xx (unit) | |
| | | | | Monocytes | xx (unit) H | |
| | | | | Other: xxxxx | xx (unit) | |
| | Baseline Visit 1b | ddmmmyyyy/ | Xxxxxxxxxxx/<br>xxxxxxx | WBC | xx (unit) | Xx |
| | | AA | ΑΛΑΛΑΛ | Hemoglobin | xx (unit) | Xx |

L=Low and H=High relative to normal ranges.

Day is calculated relative to the day of first dose of study medication.


Listing 16.3-2.1 (page 1 of n)
Blood Chemistry by Visit
All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Sample<br>Date/ Day | Laboratory<br>Number / Name | Parameter | Result (units) | CTC Grade |
|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit | ddmmmyyyy/<br>xx | Xxxxxxxxxx/<br>xxxxxxxxxxx | Urea | xx (unit) | |
| | | | | BUN | xx (unit) | |
| | | | | Creatinine | xx (unit) L | Xx |
| | | | | LDH | xx (unit) L | |
| | | | | Total Protein | xx (unit) L | |
| | | | | Albumin | xx (unit) | Xx |
| | | | | Total Bilirubin | xx (unit) | Xx |
| | | | | SGOT (AST) | xx (unit) | Xx |
| | | | | SGPT (ALT) | xx (unit) | Xx |
| | | | | Alkaline | xx (unit) | Xx |
| | | | | Phosphatase | (41120) | |
| | Baseline Visit 1b | ddmmmyyyy/<br>xx | Xxxxxxxxxx/<br>xxxxxxxxxxx | Urea | xx (unit) | |
| | | | | BUN | xx (unit) | |

L=Low and H=High relative to normal ranges.

Day is calculated relative to the day of first dose of study medication.


Listing 16.3-3.1 (page 1 of n) Serum Lipid Profile by Visit All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Sample<br>Date/ Day | Laboratory<br>Number / Name | Parameter | Result<br>(units) | CTC<br>Grade |
|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit<br>1a | ddmmmyyyy/<br>xx | Xxxxxxxxxx/<br>xxxxxxxxxxx | Total<br>Cholesterol<br>Triglycerides<br>LDL<br>HDL | xx (unit) xx (unit) xx (unit) L xx (unit) L xx (unit) L | Xx<br>Xx |
| | Baseline Visit 1b | ddmmmyyyy/<br>xx | Xxxxxxxxx/<br>xxxxxxxxxxx | Total<br>Cholesterol<br>Triglycerides | xx (unit) xx (unit) | xx |

L=Low and H=High relative to normal ranges.

Day is calculated relative to the day of first dose of study medication.


Listing 16.3-4.1 (page 1 of n)
Coagulation by Visit
All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Sample<br>Date/ Day | Laboratory<br>Number / Name | Parameter | Result<br>(units) |
|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit | ddmmmyyyy/<br>xx | Xxxxxxxxxx/<br>xxxxxxxxxxx | PT | xx (unit) |
| | 1a | ** | ********* | INR | xx (unit) L |
| | Cycle 2 Visit 4 | ddmmmyyyy/ | Xxxxxxxxxx/ | PT | xx (unit) L |
| | | XX | xxxxxxxxxx | INR | XX |

L=Low and H=High relative to normal ranges.

Day is calculated relative to the day of first dose of study medication.


Listing 16.3-5.1 (page 1 of n)
Urinalysis Dipstick Analysis by Visit
All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Sample<br>Date/ Day | Laboratory<br>Number / Name | Parameter | Result |
|---|---|---|---|---|---|
| Xxxxxxxxxx/ | Screening Visit | ddmmmyyyy/ | Xxxxxxxxxx/ | Specific | Xx |
| Xxxx-xxxxx | 1a | XX | xxxxxxxxxx | Gravity | |
| | | | | рН | Xx L |
| | | | | Protein | Xx |
| | | | | Glucose | Xx |
| | | | | Bilirubin | Xx |
| | | | | Ketones | Xx |
| | | | | Blood Cells | Xx |
| | | | | Leukocytes | Xx |
| Xxxxxxxxxx/ | Screening Visit | ddmmmyyyy/ | Xxxxxxxxxx/ | Specific | Xx L |
| Xxxx-xxxx | 1a | XX | XXXXXXXXXX | Gravity | |
| | | | | рН | Xx |
| | | | | Protein | Xx |
| | | | | Glucose | Xx |
| | | | | Bilirubin | Xx |
| | | | | Ketones | Xx |
| | | | | Blood Cells | Xx |
| | | | | Leukocytes | Xx |

L=Low and H=High relative to normal ranges.

Day is calculated relative to the day of first dose of study medication.


## Listing 16.3-5.2 (page 1 of n) Urinalysis Microscopic Analysis by Visit All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Sample<br>Date/ Day | Any Abnormal<br>Results | Sample Name | Result | Value |
|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit<br>1a | ddmmmyyyy/<br>xx | No | | | |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit<br>1a | ddmmmyyyy/<br>xx | No | | | |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Screening Visit<br>1a | ddmmmyyyy/<br>xx | Yes | UWBC/HPF<br>Present<br>Casts/LPF<br>Present | Not Present Present | xxxx |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then by visit date. Any abnormal results will be sorted by the order they appear on the CRF.


## Listing 16.4-1.1 (page 1 of n) Concomitant Medications and Non-Drug Therapies All Treated Patients

| Country/ | ATC Class/ | | | | | | |
|---|---|---|---|---|---|---|---|
| Centre/ | Preferred Term/ | | | | | Start Date/ | End Date/ |
| Patient | Medication or Non-Drug Therapy | Dose | Frequency | Route | Reason | Day | Day |
| Xxxxxxxxxx/ | Xxxxxxxxxx/ | Xx mg | 2x daily | PO | xxxxxxxxxxx | ddmmmyyyy/ | ddmmmyyyy/ |
| Xxxx-xxxxx | Xxxxxxxxxxxxx ^ | _ | - | | | XX | XX |
| | Xxxxxxxxxxx/ | Xx mg | Xxxxxx | Nasal | xxxxxxxxxx | ddmmmyyyy/ | ddmmmyyyy/ |
| | Xxxxxxxxxxxxx | | | | | XX | XX |
| | Xxxxxxxxxxx/ | Xx | On demand | Other | XXXXXXXXXX | ddmmmyyyy/ | ddmmmyyyy/ |
| | Xxxxxxxxxxxx | patch | | | | XX | XX |
| | Xxxxxxxxxxx/ | Xx mg | 1x weekly | Oral | XXXXXXXXXX | ddmmmyyyy/ | Ongoing |
| | Xxxxxxxxxxxx | | | | | XX | |
| Xxxxxxxxxx/ | Xxxxxxxxxx/ | Xx mq | 2x daily | PO | xxxxxxxxxxx | ddmmmyyyy/ | Ongoing |
| Xxxx-xxxxx | Xxxxxxxxxxxxxx ^ | _ | - | | | XX | , |
| | Xxxxxxxxxxx/ | Xx mg | Xxxxxx | Nasal | xxxxxxxxxx | ddmmmyyyy/ | ddmmmyyyy/ |
| | xxxxxxxxxxxx | | | | | XX | XX |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then by medications/therapies in order of start date (oldest first). Where unit or frequency have been recorded as "other" and then specified, it is only necessary to show the text in the specification (rather than Other: xxxxx). For route it appears from the CRF design that there is no further specification if "Other" is recorded so in this case the listing should just present "Other".

<sup>^</sup> Prior Medication


## Listing 16.4-2.1 (page 1 of n) Antineoplastic Therapy Since Discontinuation of Study Drug All Treated Patients

| Country/<br>Centre/ Patient | Regimen<br>Number | Therapy Type | Medication/<br>Non-Drug<br>Therapy | Start Date/<br>Day | Stop Date/<br>Day |
|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Chemotherapy | xxxxxxxxx | ddmmmyyyy/ xx | Ongoing |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Immunotherapy | xxxxxxxxx | ddmmmyyyy/ xx | ddmmmyyyy/ xx |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | 1 | Other:<br>xxxxxxxx | xxxxxxxx | ddmmmyyyy/ xx | ddmmmyyyy/ xx |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier. Therapy should be ordered by Regimen Number.


Listing 16.5-1.1 (page 1 of n)
All Adverse Events
All Treated Patients

| Country/<br>Centre/<br>Patient | System Organ Class/<br>Preferred Term/<br>Verbatim | Serious<br>Adverse<br>Event | Grade | Relationship<br>Suspected? /<br>Action Taken | Resulted in Death? | Start Date/<br>Day | End Date/<br>Day | Treatment<br>Emergent<br>Event |
|---|---|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Xxxxxxxxxxx/<br>Xxxxxxxxxxxxx/ | Yes | 4 | No/<br>No Action Taken | No | ddmmmyyyy/<br>xx | ddmmmyyyy/<br>xx | No |
| | Xxxxxxxxx<br>Xxxxxxxxxxxx/<br>Xxxxxxxxxxxxxxx | No | 2 | No/<br>Conmed Given | No | ddmmmyyyy/<br>xx | ddmmmyyyy/<br>xx | Yes |
| | Xxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxxxx | No | 1 | Yes/<br>Temporarily stopped<br>study drug | No | ddmmmyyyy/<br>xx | ddmmmyyyy/<br>xx | Yes |
| | Xxxxxxxxxxx/<br>Xxxxxxxxxxxxx/<br>xxxxxxxxxx | No | 1 | No/<br>No action taken | No | ddmmmyyyy/<br>xx | Ongoing | Yes |
| Xxxxxxxxx/<br>Xxxx-xxxxx | Xxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxx | No | 2 | No/<br>Permanently stopped<br>study drug | Yes | ddmmmyyyy/<br>xx | ddmmmyyyy/<br>xx | No |

Day is calculated relative to the day of first dose of study medication.

Adverse events are flagged as resulting in death if the patient dies and the AE end date is the day of death or is missing.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then by adverse event in order of start date (oldest first).

The following listings will follow this format: Listing 16.5-2.1 Deaths Reportable as SAEs - All Patients Listing 16.5-2.2 Non-Fatal SAEs - All Patients


Listing 16.6-1.1 (page 1 of n)
RECIST Solid Tumor Response Assessment - Target Lesions
All Treated Patients

| Country/<br>Centre/ | | Visit Date/ | Lesion | | Evaluation | Date of<br>Baseline | Baseline<br>Evaluation | Date of<br>Evaluation | Evaluation |
|---|---|---|---|---|---|---|---|---|---|
| Patient | Visit | Day | Number | Location | Method | Evaluation | Method | 1 | 1 (mm) |
| - | | _ | | | | | | | |
| Xxxxxxxxxx/ | Cycle 3 | ddmmmyyyy/ | 1 | XXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| Xxxx-xxxxx | Visit 7 | XX | | | | | | | |
| | | | 2 | XXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| | Cycle 6 | ddmmmyyyy/ | 1 | XXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| | Visit 10 | XX | | | | | | | |
| | | | 2 | XXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| | Cycle 9 | ddmmmyyyy/ | 1 | XXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| | Visit 13 | XX | | | | | | | |
| | | | 2 | XXXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| | Cycle 12 | ddmmmyyyy/ | 1 | XXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| | Visit 16 | XX | | | | | | | |
| | | | 2 | XXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| | Cycle 15 | ddmmmyyyy/ | 1 | XXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |
| | Visit 19 | XX | | | | | | | |
| | | | 2 | XXXXXXXX | 4 | ddmmmyyyy | 4 | ddmmmyyyy | XX.X |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then visit. Lesions should be sorted by Lesion Number. Any unscheduled assessments should be included and labeled "Unscheduled Visit".


Listing 16.6-1.2 (page 1 of n)

RECIST Solid Tumor Response Assessment - Non-Target Lesions

All Treated Patients

| Country/<br>Centre/<br>Patient | Visit | Visit Date/<br>Day | Lesion<br>Number | Location | Evaluation<br>Method | Date of<br>Baseline<br>Evaluation | Baseline<br>Evaluation<br>Method | Date of<br>Evaluation<br>1 | Evaluation<br>1 |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | _ | | _ | | |
| Xxxxxxxxxx/ | Cycle 3 | ddmmmyyyy/ | 1 | XXXXXXXX | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxx |
| Xxxx-xxxxx | Visit 7 | XX | | | | | | | |
| | | | 2 | XXXXXXXX | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxx |
| | Cycle 6 | ddmmmyyyy/ | 1 | XXXXXXX | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxx |
| | Visit 10 | XX | | | | | | | |
| | | | 2 | xxxxxxx | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxx |
| | Cycle 9 | ddmmmyyyy/ | 1 | xxxxxxx | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxxx |
| | Visit 13 | XX | | | | 1111 | | | |
| | | | 2 | xxxxxxx | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxx |
| | Cycle 12 | ddmmmyyyy/ | 1 | XXXXXXXX | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxxx |
| | Visit 16 | XX | - | *************************************** | • | admining f f f | • | • | *************************************** |
| | V1510 10 | AA | 2 | xxxxxxxx | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxxx |
| | 0115 | 1.1/ | | | | | | | |
| | Cycle 15 | ddmmmyyyy/ | 1 | XXXXXXX | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxx |
| | Visit 19 | XX | | | | | | | |
| | | | 2 | XXXXXXXX | 4 | ddmmmyyyy | 4 | 4 | Xxxxxxx |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then visit. Lesions should be sorted by Lesion Number. Any unscheduled assessments should be included and labeled "Unscheduled Visit".


Listing 16.6-1.3 (page 1 of n)
RECIST Solid Tumor Response Assessment - Overall Response
All Treated Patients

| Country/ | | | | | Overall |
|-------------|----------|-------------|------------|-----------|----------|
| Centre/ | | Visit Date/ | Evaluation | Date of | Lesion |
| Patient | Visit | Day | Number | Response | Response |
| Xxxxxxxxxx/ | Cycle 3 | ddmmmyyyy/ | 1 | ddmmmyyyy | Xxxxxxx |
| Xxxx-xxxxx | Visit 7 | XX | | | |
| | | | 2 | ddmmmyyyy | Xxxxxxx |
| | Cycle 6 | ddmmmyyyy/ | 1 | ddmmmyyyy | Xxxxxxx |
| | Visit 10 | XX | | | |
| | | | 2 | ddmmmyyyy | Xxxxxxxx |
| | Cycle 9 | ddmmmyyyy/ | 1 | ddmmmyyyy | Xxxxxxxx |
| | Visit 13 | XX | | | |
| | | | 2 | ddmmmyyyy | Xxxxxxx |
| | Cycle 12 | ddmmmyyyy/ | 1 | ddmmmyyyy | Xxxxxxx |
| | Visit 16 | XX | | | |
| | | | 2 | ddmmmyyyy | Xxxxxxx |
| | Cycle 15 | ddmmmyyyy/ | 1 | ddmmmyyyy | Xxxxxxxx |
| | Visit 19 | XX | | 2222 | |
| | | | 2 | ddmmmyyyy | Xxxxxxx |
| | | | 2 | ddmmmyyyy | Xxxxxxx |

Day is calculated relative to the day of first dose of study medication.

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then visit. Evaluations should be sorted by Evaluation Number. Any unscheduled assessments should be included and labeled "Unscheduled Visit".


Listing 16.6-1.4 (page 1 of n)
Survival Status at End of Study
All Treated Patients

| Country/<br>Centre/ | Current | Death Date/ | | Last Contact<br>Date/ |
|---|---|---|---|---|
| Patient | Status | Day | Principal Cause of Death | Day |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Alive | | | ddmmmyyyy/<br>xx |
| Xxxxxxxxxx/ | Lost to | | | ddmmmyyyy/ |
| Xxxx-xxxxx | Follow-up | | | xx |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Dead | ddmmmyyyy/<br>xx | Other: xxxxxxxxxxxxxxxxxxxxxxxx | |
| Xxxxxxxxxx/ | Alive | | | ddmmmyyyy/ |
| Xxxx-xxxxx | | | | xx |
| Xxxxxxxxxx/ | Dead | ddmmmyyyy/ | Study Indication | |
| Xxxx-xxxxx | | XX | | |

Day is calculated relative to the day of first dose of study medication.


Listing 16.6-1.5 (page 1 of n)
Progression and Survival Details
All Treated Patients

| Country/<br>Centre/<br>Patient | Progression<br>Status | Date of<br>First<br>Progression<br>Event | Days from<br>Start of<br>Treatment to<br>Progression | Survival<br>Status | Date of<br>Death/<br>Last<br>Contact | Days from<br>Start of<br>Treatment<br>to Death | Disease<br>Control | Objectiv<br>e<br>Response | Duration<br>of<br>Response<br>(Days) |
|---|---|---|---|---|---|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Progression | ddmmmyyyy | xx | Dead | ddmmmyyyy | xx | No | No | |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | No<br>Progression | ddmmmyyyy | xx^ | Alive | ddmmmyyyy | xx^ | Yes | Yes | xx |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Progression | ddmmmyyyy | XX | Alive | ddmmmyyyy | xx^ | No | No | |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | No<br>Progression | ddmmmyyyy | xx^ | Alive | ddmmmyyyy | XX^ | Yes | Yes | xx^ |

<sup>^</sup>Censored


Listing 16.7-1.1 (page 1 of n)
Comments Listing
All Patients

| Country/<br>Centre/<br>Patient | Cycle | Page Number | Comments |
|---|---|---|---|
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Cycle 1 | Xxx | Xxxxxxx xxxxxxx xxxxx xxxxxxxxxxxxxxxx |
| | Cycle 4 | Xxx | Xxxxxxxxx xxxxxxxxx xxxxxxxxxxx xxxxxxxx |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | Cycle 2 | Xxx | Xxxxxxxxx xxxxxxxxx xxxxxxxx xxxxxxxx |
| Xxxxxxxxxx/<br>Xxxx-xxxxx | End of<br>Treatment | Xx | Xxxxxxxxx xxxxxxxxx xxxxxxxx |

Programming note: Data ordered by country (alphabetically) then centre/patient identifier then by cycle and page number.